CLINICAL TRIAL: NCT02801942
Title: Exploration of the Peripheral Immune System in Subjects With New Onset T1 Diabetes (NOT1D)
Brief Title: Immune Profile in Subjects With New Onset Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 203158
Record Dates: First submitted 2016-06-13; First posted 2016-06-16 (Estimated); Results first posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2018-07

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Biomarker; Immune Profile; Biopsy; Leukocyte subsets; Inguinal lymph nodes; Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Lead

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy subjects (Experimental): Up to 30 mL of blood sample will be collected from healthy subjects. Inguinal lymph node fine needle aspirate biopsy and core biopsy will be performed. Leukocyte subset phenotyping will be carried out on iLN-derived cells by assessing expression of (but not restricted to) the following antigens: CD3, CD4, CD8, CD11c, CD14, CD16, CD19, CD24, CD25, CD38, CD45RA, CD56, Human Leukocyte antigen D related (HLA-DR) and forkhead box P3 protein also called scurfin (FOXP3).
  Interventions: Procedure: Inguinal lymph node fine needle aspirate biopsy; Procedure: Inguinal lymph node core biopsy; Procedure: Peripheral blood collection; Other: Pre- and post-biopsy questionnaire
- Subjects with NOT1D (Experimental): Up to 30 mL of blood sample will be collected from subjects with NOT1D. Inguinal lymph node fine needle aspirate biopsy and core biopsy will be performed. Leukocyte subset phenotyping will be carried out on iLN-derived cells by assessing expression of (but not restricted to) the following antigens: CD3, CD4, CD8, CD11c, CD14, CD16, CD19, CD24, CD25, CD38, CD45RA, CD56, HLA-DR and FOXP3.
  Interventions: Procedure: Inguinal lymph node fine needle aspirate biopsy; Procedure: Inguinal lymph node core biopsy; Procedure: Peripheral blood collection; Other: Pre- and post-biopsy questionnaire

INTERVENTIONS:
Procedure: Inguinal lymph node fine needle aspirate biopsy — Inguinal lymph node will be localized by ultrasonography and sampled by 21-gauge needle and a 5 mL syringe using to and fro needle movement while applying 1 mL suction with the syringe. Up to 2 fine needle aspirate passages will be obtained, to derive immune cells.
Procedure: Inguinal lymph node core biopsy — Inguinal lymph node will be localized by ultrasonography and following fine needle aspirate, an incision will be made. Up to five core biopsies will be obtained, to derive immune cells.
Procedure: Peripheral blood collection — Blood sample (30 mL) will be collected, to derive immune cells.
Other: Pre- and post-biopsy questionnaire — All subjects will be asked to complete a questionnaire about their expectations/experiences of undergoing the biopsy procedures.

SUMMARY:
It is hypothesized that early changes in the immune system in New Onset Type 1 Diabetes Mellitus (NOT1D) subjects can be detected in immune cells from the inguinal lymph nodes (iLN), which will be distinct from changes observed in peripheral blood derived immune cells. Therefore this study will assess and compare the molecular immune profile of cells derived from the iLN in healthy and NOT1D subjects, to understand the immunological processes that may lead to beta cell destruction. It is a multi-center, non-drug treatment study. Up to 15 subjects in each group, namely healthy subjects and NOT1D subjects, will be evaluated in the study. A data look will be carried out after the recruitment of a cohort of up to 5 healthy subjects, to determine if the quality and quantity of cells derived from aspirate or core biopsy or from peripheral blood are likely to be sufficient to continue the study to meet its primary objective. An interim analysis will be carried out after the recruitment of 5 evaluable healthy subjects and 5 evaluable NOT1D subjects. The primary purpose of this interim analysis will be to facilitate decision making and study design for a potential follow-up interventional study.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 40 years of age inclusive, at the time of signing the informed consent.
* Healthy subjects will be as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination and laboratory tests.
* Subjects will be considered healthy if values for the following parameters: fasted glucose, glycated hemoglobin (HbA1c), International normalized ratio (INR), activated partial thromboplastin time (APTT), platelet count, red blood cells and total lymphocyte count are within the normal range at screening.
* NOT1D subject with documented diagnosis of diabetes mellitus according to American Diabetes Association (ADA) and World Health Organization (WHO) criteria and consistent with Type 1a (autoimmune) Diabetes Mellitus, with an interval of up to 8 weeks between the initial diagnosis and day 1 of the study (Day 1 = "iLN biopsy" day).
* NOT1D subject, who currently requires insulin treatment for type 1 diabetes (T1D) and has received insulin therapy for at least 7 days prior to screening.
* NOT1D subject positive, at screening, for at least one autoantibody associated with T1D: anti- Glutamic Acid Decarboxylase (GAD), anti-Islet antigen 2 (IA-2), anti- islet cell antibodies (ICA), anti-Indole 3 acetic acid (IAA), anti- Zinc transporter 8 (ZnT8).
* NOT1D subject with evidence, at screening, of residual functioning beta cells as measured by fasted C-peptide levels >=0.15 nanomole per liter (nmol/L).
* NOT1D subject having values for the following parameters: INR, APTT, platelet count, red blood cells and total lymphocyte count within the normal range at screening.
* Both, male or female subjects are eligible to participate in this study. A female subject is only eligible to participate if she is not pregnant [as confirmed by a negative urine human chorionic gonadotropin (hCG) test], not lactating at screening and study visit(s) or has documented evidence to not be of child bearing potential.
* Capable of giving signed informed consent which includes compliance with the study requirements and study restrictions.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator, in consultation with the Medical Monitor if required, agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.

Exclusion Criteria:

* Healthy subjects having family history of T1D (that is, first degree relative has been diagnosed with T1D)
* Healthy subjects with presence of one or more of serum autoantibodies, such as anti-GAD, anti-IA2, anti-ICA, anti-IAA, anti-ZnT8, anti-thyroid peroxidase antibodies, anti-tissue transglutaminase antibodies and anti-nuclear antibodies.
* NOT1D subjects with history of autoimmune disease other than T1D
* NOT1D subjects with presence of one or more of serum autoantibodies of the following: anti-thyroid peroxidase antibodies, anti-tissue transglutaminase antibodies or anti-nuclear antibodies
* Allergy or intolerance to local anesthetic agents
* Any localized groin condition which would contraindicate biopsy procedure including but not limited to: Active infection/inflammation at the intended puncture site, previous surgery/scarring or any other anatomical abnormality as deemed relevant to the procedure by the investigator, in consultation with the Medical Monitor if required.
* History of bleeding disorders, current or anticipated continuous use of anticoagulant (including but not limited to warfarin, rivaroxaban) and antiplatelet agents (including but not limited to Nonsteroidal anti-inflammatory drugs [NSAIDS], clopidogrel, etc.)
* Active or unresolved bacterial infection, viral infection, fungal infection within 4 weeks prior to day 1.
* Known febrile episode over 38 degrees Celsius within 4 weeks prior to day 1.
* Active organ dysfunction or previous organ allograft.
* History of malignancy (with the exception of resected basal carcinoma of the skin or cervical carcinoma in situ).
* Has undergone any major surgical procedure within 30 days before screening, and/or is planning to undergo any such surgery during the period of the study (i.e. from screening until the last follow-up telephone call)
* Present or previous treatment with any cell depleting therapies or immune-modulating or suppressive agents (e.g., oral steroids), including investigational agents such as the following but not limited to e.g., Interleukin (IL)-2, alemtuzumab, anti- Cluster of Differentiation (CD) 4, anti-CD5, anti-CD3, anti-CD19, anti-CD20.
* Vaccination =<28 days before day 1 of the study or planned during the study period
* Current participation in an interventional clinical trial. Subjects, who participated in an interventional clinical trial previously, must wait for 3 months after completing the previous interventional clinical trial before participating in this study.
* Any medical history or clinically relevant abnormality that is deemed by the investigator and/or medical monitor to make the subject ineligible for inclusion because of a safety concern or any situation that, in the investigator's judgment, is likely to cause the subject to be unable or unwilling to participate in study procedures or to complete all scheduled assessments.
* A positive pre-study drug/alcohol screen (unless positive due to prescription medication). A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* Inability to access the groin area to perform the biopsy procedure as judged by the investigator.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2016-07-25 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United Kingdom (2):
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, Cardiff

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multi-center, non-drug treatment study to compare differences in immune cells derived from the inguinal lymph nodes (iLN) and peripheral blood of New Onset Type 1 Diabetes Mellitus (NOT1D) participants and healthy volunteers. Participants were enrolled at a single center in United Kingdom.
Pre-assignment Details: Participants underwent iLN biopsies by two methods; fine-needle aspirate (FNA) and core needle biopsy. Participants underwent screening followed by study visits and follow-up. A total of 43 participants were screened, of which, 21 were considered as screen failures and 22 were enrolled into the study.
Groups:
- Healthy Participants: Participants were considered healthy if values for the following parameters: fasted glucose, glycated hemoglobin, International normalized ratio (INR), activated partial thromboplastin time (APTT), platelet count, red blood cells and total lymphocyte count were within the normal range at screening.
- Participants With NOT1D: NOT1D participants with documented diagnosis of diabetes mellitus according to American Diabetes Association (ADA) and World Health Organization (WHO) criteria and consistent with Type 1a (autoimmune) Diabetes Mellitus, were included in the study.
Period: Overall Study
Arm/Group | Healthy Participants | Participants With NOT1D
Started | 12 | 10
Completed | 12 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Participants | Participants With NOT1D | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.6 (5.53) | 27.0 (5.35) | 27.9 (5.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 8 | 6 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - White/Caucasian/European Heritage | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Leukocyte Subsets Including B Lymphocytes, Classical B Lymphocytes, Double Negative B Lymphocytes, Naive B Lymphocytes, Plasmablast and Transitional B Lymphocytes in Blood
Description: Peripheral blood samples were collected from both healthy and NOT1D participants at the indicated time points for the analysis of leukocyte subsets from Monocyte Panel. Candidate biomarkers associated with either location of cells and/or disease-status were identified using flow cytometry technique. Generalized linear mixed models were used to analyze data separately for each flow cytometry cell type to provide estimates for comparisons. Fixed categorical were group, sample type, and the interaction of group with sample type, where Group was HV or NOT1D, and sample type was peripheral blood, core biopsy or FNA. The analysis was based upon Safety Population which comprised of all participants who complete any study assessment. Only those participants with data available at specific time point were analyzed (represented by n=x in category titles). NA indicates that data was not available.
Time Frame: Pre Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of B lymphocytes
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of B lymphocytes
  Circulating B Lymphocytes; n=12, 10 | 16.54 (2.229) | 14.23 (2.442)
  Classical B Lymphocytes; n=12, 10 | 19.37 (1.616) | 15.83 (1.771)
  Double Negative B Lymphocytes; n=12, 10 | 3.25 (1.250) | 6.26 (1.370)
  Naive B Lymphocytes; n=12, 10 | 59.81 (3.021) | 62.32 (3.310)
  Plasmablast ; n=11, 10: number analyzed (Participants) | 11 | 10
  Plasmablast ; n=11, 10 | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis. | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.
  Transitional B Lymphocytes; n=12, 10 | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis. | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 2.31, 95% CI 2-sided [-4.59 to 9.21], Standard Error of Mean 3.307 — The mean difference in circulating B lymphocytes (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 3.54, 95% CI 2-sided [-1.46 to 8.54], Standard Error of Mean 2.398 — The mean difference in Classical B Lymphocytes (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -3.01, 95% CI 2-sided [-6.87 to 0.86], Standard Error of Mean 1.854 — The mean difference in Double Negative B Lymphocytes (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 4: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -2.51, 95% CI [-11.86 to 6.84], Standard Error of Mean 4.482 — The mean difference in Naive B Lymphocytes (Healthy participants versus NOT1D participants) in blood has been presented

2. Primary Outcome: Percentage of Leukocyte Subsets Including B Lymphocytes, Classical B Lymphocytes, Double Negative B Lymphocytes, Naive B Lymphocytes, Plasmablast and Transitional B Lymphocytes in iLN
Description: Samples were collected including up to two FNA passages of iLN and up to five core biopsies of iLN at the indicated time point from both healthy and NOT1D participants for the analysis of leukocyte subsets from Monocyte Panel. Candidate biomarkers associated with either location of cells and/or disease-status were identified using flow cytometry technique. Generalized linear mixed models were used to analyze data separately for each flow cytometry cell type to provide estimates for comparisons. Fixed categorical were group, sample type, and the interaction of group with sample type, where Group was HV or NOT1D, and sample type was peripheral blood, core biopsy or FNA. Only those participants with data available at specific time point were analyzed (represented by n=x in category titles). NA indicates that data was not available.
Time Frame: Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of B lymphocytes
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of B lymphocytes
  Circulating B Lymphocytes; n=9, 10: number analyzed (Participants) | 9 | 10
  Circulating B Lymphocytes; n=9, 10 | 15.51 (1.860) | 12.14 (1.898)
  Classical B Lymphocytes; n=9, 10: number analyzed (Participants) | 9 | 10
  Classical B Lymphocytes; n=9, 10 | 38.78 (4.119) | 30.19 (4.130)
  Double Negative B Lymphocytes; n=9, 10: number analyzed (Participants) | 9 | 10
  Double Negative B Lymphocytes; n=9, 10 | 8.68 (1.668) | 10.26 (1.651)
  Naive B Lymphocytes; n=9, 10: number analyzed (Participants) | 9 | 10
  Naive B Lymphocytes; n=9, 10 | 35.83 (3.761) | 44.13 (3.621)
  Plasmablast; n=4, 8: number analyzed (Participants) | 4 | 8
  Plasmablast; n=4, 8 | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis. | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.
  Transitional B Lymphocytes; ; n=3, 2: number analyzed (Participants) | 3 | 2
  Transitional B Lymphocytes; ; n=3, 2 | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis. | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 3.38, 95% CI 2-sided [-2.22 to 8.98], Standard Error of Mean 2.658 — The mean difference in Circulating B Lymphocytes (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 8.59, 95% CI 2-sided [-3.72 to 20.91], Standard Error of Mean 5.833 — The mean difference in Classical B Lymphocytes (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -1.58, 95% CI 2-sided [-6.53 to 3.38], Standard Error of Mean 2.347 — The mean difference in Double Negative B Lymphocytes (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 4: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -8.31, 95% CI 2-sided [-19.32 to 2.71], Standard Error of Mean 5.221 — The mean difference in Naive B Lymphocytes (Healthy participants versus NOT1D participants) in iLN has been presented

3. Primary Outcome: Percentage of Leukocyte Subsets Including B-cells, Clusters of Differentiation 56 Positive (CD56+) CD16+ , CD56bright Natural Killer (NK) Cells, CD56lo CD16+, CD56lo CD16 Negative (CD56lo CD16-), Dendritic Cells, NK Cells in Blood
Description: Peripheral blood samples were collected from both healthy and NOT1D participants at the indicated time points for the analysis of leukocyte subsets from Monocyte Panel. Candidate biomarkers associated with either location of cells and/or disease-status were identified using flow cytometry technique. Generalized linear mixed models were used to analyze data separately for each flow cytometry cell type to provide estimates for comparisons. Fixed categorical were group, sample type, and the interaction of group with sample type, where Group was HV or NOT1D, and sample type was peripheral blood, core biopsy or FNA. NA indicates that data was not available.
Time Frame: Pre Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of mononuclear cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of mononuclear cells
  B-cells | 8.50 (0.589) | 7.58 (0.645)
  CD56+CD16+ | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis. | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.
  CD56bright NK cells | 0.36 (0.042) | 0.30 (0.046)
  CD56lo CD16+ | 7.96 (1.011) | 8.24 (1.108)
  CD56lo CD16- | 0.24 (0.036) | 0.23 (0.040)
  Dendritic cells | 0.93 (0.080) | 0.87 (0.088)
  NK cells | 8.71 (0.999) | 8.84 (1.095)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.92, 95% CI 2-sided [-0.90 to 2.75], Standard Error of Mean 0.873 — The mean difference in B-cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.07 to 0.19], Standard Error of Mean 0.063 — The mean difference in CD56bright NK cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-3.41 to 2.84], Standard Error of Mean 1.500 — The mean difference in CD56lo CD16+ (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 4: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.10 to 0.13], Standard Error of Mean 0.054 — The mean difference in CD56lo CD16- (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 5: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.19 to 0.31], Standard Error of Mean 0.118 — The mean difference in Dendritic cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 6: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-3.23 to 2.96], Standard Error of Mean 1.482 — The mean difference in NK cells (Healthy participants versus NOT1D participants) in blood has been presented

4. Primary Outcome: Percentage of Leukocyte Subsets Including B-cells, CD56+ CD16+, CD56bright NK Cells, CD56lo CD16+, CD56lo CD16-, Dendritic Cells, NK Cells in iLN
Description: as for outcome 2
Time Frame: Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of mononuclear cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of mononuclear cells
  B-cells; n=9, 10: number analyzed (Participants) | 9 | 10
  B-cells; n=9, 10 | 8.88 (1.641) | 7.34 (1.512)
  CD56+CD16+; n=8, 8: number analyzed (Participants) | 8 | 8
  CD56+CD16+; n=8, 8 | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis. | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.
  CD56bright NK cells; n=9, 10: number analyzed (Participants) | 9 | 10
  CD56bright NK cells; n=9, 10 | 0.54 (0.098) | 0.50 (0.101)
  CD56lo CD16+; n=9, 10: number analyzed (Participants) | 9 | 10
  CD56lo CD16+; n=9, 10 | 0.68 (0.173) | 0.69 (0.184)
  CD56lo CD16-; n=8, 9: number analyzed (Participants) | 8 | 9
  CD56lo CD16-; n=8, 9 | 0.19 (0.043) | 0.21 (0.040)
  Dendritic cells; n=9, 10: number analyzed (Participants) | 9 | 10
  Dendritic cells; n=9, 10 | 0.45 (0.100) | 0.39 (0.081)
  NK cells; n=9, 10: number analyzed (Participants) | 9 | 10
  NK cells; n=9, 10 | 1.43 (0.324) | 1.50 (0.364)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 1.54, 95% CI 2-sided [-3.14 to 6.23], Standard Error of Mean 2.231 — The mean difference in B-cells in (Healthy participants versus NOT1D participants) iLN has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.25 to 0.34], Standard Error of Mean 0.140 — The mean difference in CD56bright sNK cells (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.54 to 0.52], Standard Error of Mean 0.253 — The mean difference in CD56lo CD16+ (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 4: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.15 to 0.10], Standard Error of Mean 0.059 — The mean difference in CD56lo CD16- (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 5: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.21 to 0.34], Standard Error of Mean 0.128 — The mean difference in Dendritic cells (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 6: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-1.10 to 0.96], Standard Error of Mean 0.487 — The mean difference in NK cells (Healthy participants versus NOT1D participants) in iLN has been presented

5. Primary Outcome: Percentage of Leukocyte Subsets Including CD56+CD16+, CD56bright NK Cells, CD56lo CD16+ and CD56lo CD16- in Blood
Description: as for outcome 3
Time Frame: Pre Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of NK cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of NK cells
  CD56+CD16+ | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis. | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.
  CD56bright NK cells | 5.02 (0.894) | 3.99 (0.980)
  CD56lo CD16+ | 89.71 (1.567) | 92.40 (1.717)
  CD56lo CD16- | 3.11 (0.497) | 2.70 (0.545)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 1.03, 95% CI 2-sided [-1.73 to 3.80], Standard Error of Mean 1.326 — The mean difference in CD56bright NK cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -2.69, 95% CI 2-sided [-7.54 to 2.16], Standard Error of Mean 2.324 — The mean difference in CD56lo CD16+ (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.42, 95% CI 2-sided [-1.12 to 1.95], Standard Error of Mean 0.738 — The mean difference in CD56lo CD16- (Healthy participants versus NOT1D participants) in blood has been presented

6. Primary Outcome: Percentage of Leukocyte Subsets Including CD56+CD16+, CD56bright NK Cells CD56lo CD16+ and CD56lo CD16- in iLN
Description: as for outcome 2
Time Frame: Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of NK cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of NK cells
  CD56+CD16+; n=8, 8: number analyzed (Participants) | 8 | 8
  CD56+CD16+; n=8, 8 | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis. | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.
  CD56bright NK cells; n=9, 10: number analyzed (Participants) | 9 | 10
  CD56bright NK cells; n=9, 10 | 41.85 (3.999) | 35.01 (3.868)
  CD56lo CD16+; n=9, 10: number analyzed (Participants) | 9 | 10
  CD56lo CD16+; n=9, 10 | 37.12 (6.220) | 45.01 (4.900)
  CD56lo CD16-; n=8, 9: number analyzed (Participants) | 8 | 9
  CD56lo CD16-; n=8, 9 | 12.80 (1.855) | 14.26 (1.490)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 6.84, 95% CI 2-sided [-4.92 to 18.60], Standard Error of Mean 5.564 — The mean difference in CD56bright NK cells (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -7.89, 95% CI 2-sided [-24.77 to 9.00], Standard Error of Mean 7.918 — The mean difference in CD56lo CD16+ (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -1.46, 95% CI 2-sided [-6.66 to 3.73], Standard Error of Mean 2.379 — The mean difference in CD56lo CD16- (Healthy participants versus NOT1D participants) in iLN has been presented

7. Primary Outcome: Percentage of Leukocyte Subsets Including Myeloid Dendritic Cells and Plasmacytoid Dendritic Cells in Blood
Description: Peripheral blood samples were collected from both healthy and NOT1D participants at the indicated time points for the analysis of leukocyte subsets from Monocyte Panel. Candidate biomarkers associated with either location of cells and/or disease-status were identified using flow cytometry technique. Generalized linear mixed models were used to analyze data separately for each flow cytometry cell type to provide estimates for comparisons. Fixed categorical were group, sample type, and the interaction of group with sample type, where Group was HV or NOT1D, and sample type was peripheral blood, core biopsy or FNA.
Time Frame: Pre Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of total dendritic cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of total dendritic cells
  Myeloid Dendritic cells | 51.78 (3.073) | 50.45 (3.366)
  Plasmacytoid Dendritic cells | 45.51 (3.140) | 47.36 (3.440)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 1.33, 95% CI 2-sided [-8.17 to 10.84], Standard Error of Mean 4.558 — The mean difference in myeloid dendritic cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -1.85, 95% CI 2-sided [-11.57 to 7.86], Standard Error of Mean 4.658 — The mean difference in plasmacytoid dendritic cells (Healthy participants versus NOT1D participants) in blood has been presented

8. Primary Outcome: Percentage of Leukocyte Subsets Including Myeloid Dendritic Cells and Plasmacytoid Dendritic Cells in iLN
Description: Samples were collected including up to two FNA passages of iLN and up to five core biopsies of iLN at the indicated time point from both healthy and NOT1D participants for the analysis of leukocyte subsets from Monocyte Panel. Candidate biomarkers associated with either location of cells and/or disease-status were identified using flow cytometry technique. Generalized linear mixed models were used to analyze data separately for each flow cytometry cell type to provide estimates for comparisons. Fixed categorical were group, sample type, and the interaction of group with sample type, where Group was HV or NOT1D, and sample type was peripheral blood, core biopsy or FNA.Only those participants with data available at specific time point were analyzed (represented by n=x in category titles).
Time Frame: Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of total dendritic cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of total dendritic cells
  Myeloid Dendritic cells; n=8, 10: number analyzed (Participants) | 8 | 10
  Myeloid Dendritic cells; n=8, 10 | 42.96 (3.870) | 30.72 (4.128)
  Plasmacytoid Dendritic cells; n=9, 9: number analyzed (Participants) | 9 | 9
  Plasmacytoid Dendritic cells; n=9, 9 | 57.43 (4.426) | 68.30 (5.372)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 12.23, 95% CI 2-sided [0.38 to 24.09], Standard Error of Mean 5.658 — The mean difference in myeloid dendritic cells (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -10.87, 95% CI 2-sided [-25.52 to 3.78], Standard Error of Mean 6.961 — The mean difference in plasmacytoid dendritic cells (Healthy participants versus NOT1D participants) in iLN has been presented

9. Primary Outcome: Percentage of Leukocyte Subsets Including CD14+ CD16+ Monocytes, CD14+ Monocytes, and CD16+ Monocytes in Blood
Description: Peripheral blood samples were collected from both healthy and NOT1D participants at the indicated time points for the analysis of leukocyte subsets from Monocyte Panel. Candidate biomarkers associated with either location of cells and/or disease-status were identified using flow cytometry technique. NA indicates that data was not available.
Time Frame: Pre Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of monocytes
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of monocytes
  CD14+ CD16+ monocytes | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis
  CD14+ monocytes | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis
  CD16+ monocytes | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis

10. Primary Outcome: Percentage of Leukocyte Subsets Including CD14+ CD16+ Monocytes, CD14+ Monocytes and CD16+ Monocytes in iLN
Description: Samples were collected including up to two FNA passages of iLN and up to five core biopsies of iLN at the indicated time point from both healthy and NOT1D participants for the analysis of leukocyte subsets from Monocyte Panel. Candidate biomarkers associated with either location of cells and/or disease-status were identified using flow cytometry technique. Only those participants with data available at specific time point were analyzed (represented by n=x in category titles). NA indicates that data was not available.
Time Frame: Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of monocytes
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of monocytes
  CD14+ CD16+ monocytes; n=0, 1: number analyzed (Participants) | 0 | 1
  CD14+ CD16+ monocytes; n=0, 1 |  | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.
  CD14+ monocytes; n=7, 4: number analyzed (Participants) | 7 | 4
  CD14+ monocytes; n=7, 4 | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis. | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.
  CD16+ monocytes; n=0, 2: number analyzed (Participants) | 0 | 2
  CD16+ monocytes; n=0, 2 |  | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.

11. Primary Outcome: Percentage of Leukocyte Subsets Including CD45RA+ Effector Memory CD8, Central Memory CD8, Effector Memory CD8, Naive CD8 and Stem Cell Memory-like CD8 Cells in Blood
Description: Peripheral blood samples were collected from both healthy and NOT1D participants at the indicated time points for the analysis of leukocyte subsets from T cell Panel. Candidate biomarkers associated with either location of cells and/or disease-status were identified using flow cytometry technique. Generalized linear mixed models were used to analyze data separately for each flow cytometry cell type to provide estimates for comparisons. Fixed categorical were group, sample type, and the interaction of group with sample type, where Group was HV or NOT1D, and sample type was peripheral blood, core biopsy or FNA.
Time Frame: Pre Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of CD8 T cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of CD8 T cells
  CD45RA+ Effector Memory CD8 | 29.89 (4.267) | 28.10 (4.674)
  Central Memory CD8 | 7.13 (1.537) | 6.98 (1.684)
  Effector Memory CD8 | 19.22 (2.223) | 14.84 (2.435)
  Naive CD8 | 34.38 (3.863) | 40.44 (4.231)
  Stem Cell Memory-like CD8 | 1.34 (0.206) | 1.37 (0.225)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 1.79, 95% CI 2-sided [-11.41 to 14.99], Standard Error of Mean 6.329 — The mean difference in CD45RA+ Effector Memory CD8 (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-4.60 to 4.91], Standard Error of Mean 2.280 — The mean difference in Central Memory CD8 (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 4.38, 95% CI 2-sided [-2.50 to 11.26], Standard Error of Mean 3.297 — The mean difference in Effector Memory CD8 (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 4: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -6.06, 95% CI 2-sided [-18.01 to 5.89], Standard Error of Mean 5.729 — The mean difference in Naive CD8 (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 5: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.67 to 0.60], Standard Error of Mean 0.305 — The mean difference in Stem Cell Memory-like CD8 (Healthy participants versus NOT1D participants) in blood has been presented

12. Primary Outcome: Percentage of Leukocyte Subsets Including CD45RA+ Effector Memory CD8, Central Memory CD8, Effector Memory CD8, Naive CD8 and Stem Cell Memory-like CD8 Cells in iLN
Description: Samples were collected including up to two FNA passages of iLN and up to five core biopsies of iLN at the indicated time point from both healthy and NOT1D participants for the analysis of leukocyte subsets from T cell Panel. Candidate biomarkers associated with either location of cells and/or disease-status were identified using flow cytometry technique. Generalized linear mixed models were used to analyze data separately for each flow cytometry cell type to provide estimates for comparisons. Fixed categorical were group, sample type, and the interaction of group with sample type, where Group was HV or NOT1D, and sample type was peripheral blood, core biopsy or FNA.
Time Frame: Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of CD8 T cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of CD8 T cells
  CD45RA+ Effector Memory CD8 | 14.54 (2.094) | 13.34 (2.330)
  Central Memory CD8 | 5.55 (0.978) | 6.21 (1.093)
  Effector Memory CD8 | 13.74 (1.867) | 15.59 (2.074)
  Naive CD8 | 55.12 (4.259) | 54.45 (4.700)
  Stem Cell Memory-like CD8 | 1.69 (0.316) | 2.36 (0.377)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 1.20, 95% CI 2-sided [-5.33 to 7.73], Standard Error of Mean 3.133 — The mean difference in CD45RA+ Effector Memory CD8 (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.66, 95% CI 2-sided [-3.73 to 2.41], Standard Error of Mean 1.466 — The mean difference in Central Memory CD8 (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -1.85, 95% CI 2-sided [-7.67 to 3.96], Standard Error of Mean 2.790 — The mean difference in Effector Memory CD8 (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 4: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.67, 95% CI 2-sided [-12.54 to 13.87], Standard Error of Mean 6.342 — The mean difference in Naive CD8 (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 5: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.67, 95% CI 2-sided [-1.71 to 0.36], Standard Error of Mean 0.492 — The mean difference in Stem Cell Memory-like CD8 (Healthy participants versus NOT1D participants) in iLN has been presented

13. Primary Outcome: Percentage of Leukocyte Subsets Including Programmed Death 1 (PD-1)+ Inducible Costimulator (ICOS)+ Follicular Helper T (TFH) Cell-like Regulatory (Reg) T Cells in Blood
Description: Peripheral blood samples were planned to be collected from both healthy and NOT1D participants at the indicated time points for the analysis of leukocyte subsets from T cell Panel. Results could not be presented as data were not collected for this analysis due to lack of model convergence or model reliability
Time Frame: Pre Biopsy session on Day 1
Population: Safety Population. Data were not collected due to lack of model convergence or model reliability.
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 0 | 0

14. Primary Outcome: Percentage of Leukocyte Subsets Including PD-1+ ICOS+ TFH Cell-like Reg T Cells in iLN
Description: Samples were collected including up to two FNA passages of iLN and up to five core biopsies of iLN at the indicated time point from both healthy and NOT1D participants for the analysis of leukocyte subsets from T cell Panel. Candidate biomarkers associated with either location of cells and/or disease-status were identified using flow cytometry technique. NA indicates that data was not available.
Time Frame: Biopsy session on Day 1
Population: Safety Population. Only those participants with data available at specified time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of TFH cell-like Reg T cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 5 | 7
Percentage of TFH cell-like Reg T cells | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis. | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.

15. Primary Outcome: Percentage of Leukocyte Subsets Including PD-1+ ICOS+ TFH Cells in Blood
Description: as for outcome 11
Time Frame: Pre Biopsy session on Day 1
Population: Safety Population. Only those participants with data available at specified time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of TFH cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 6 | 7
Percentage of TFH cells | 0.53 (0.173) | 0.87 (0.160)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-0.84 to 0.16], Standard Error of Mean 0.236 — The mean difference in PD-1+ ICOS+ TFH cells (Healthy participants versus NOT1D participants) in blood has been presented

16. Primary Outcome: Percentage of Leukocyte Subsets Including PD-1+ ICOS+ TFH Cells in iLN
Description: as for outcome 12
Time Frame: Biopsy session on Day 1
Population: Safety Population. Only those participants with data available at specified time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of TFH cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 10 | 10
Percentage of TFH cells | 2.75 (3.192) | 8.96 (2.973)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -6.21, 95% CI 2-sided [-15.37 to 2.96], Standard Error of Mean 4.362 — The mean difference in PD-1+ ICOS+ TFH cells (Healthy participants versus NOT1D participants) in iLN has been presented

17. Primary Outcome: Percentage of Leukocyte Subsets Including Central Memory Conventional (Conv) T Cells, Effector Memory Conv T Cells, Naive Conv T Cells and Stem Cell Memory-like Conv T Cells in Blood
Description: as for outcome 11
Time Frame: Pre Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of total Conv T cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of total Conv T cells
  CD45RA+ Effector Memory Conv T cells | 2.47 (0.856) | 1.44 (0.937)
  Central Memory Conv T cells | 32.21 (2.125) | 33.75 (2.328)
  Effector Memory Conv T cells | 11.74 (1.409) | 11.97 (1.543)
  Naive Conv T cells | 43.40 (2.586) | 42.48 (2.833)
  Stem Cell Memory-like Conv T cells | 0.91 (0.098) | 1.01 (0.107)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 1.03, 95% CI 2-sided [-1.61 to 3.68], Standard Error of Mean 1.269 — The mean difference in CD45RA+ Effector Memory Conv T cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -1.54, 95% CI 2-sided [-8.12 to 5.03], Standard Error of Mean 3.152 — The mean difference in Central Memory Conv T cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-4.59 to 4.13], Standard Error of Mean 2.089 — The mean difference in Effector Memory Conv T cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 4: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.92, 95% CI 2-sided [-7.08 to 8.92], Standard Error of Mean 3.835 — The mean difference in Naive Conv T cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 5: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.40 to 0.21], Standard Error of Mean 0.145 — The mean difference in Stem Cell Memory-like Conv T cells (Healthy participants versus NOT1D participants) in blood has been presented

18. Primary Outcome: Percentage of Leukocyte Subsets Including Central Memory Conv T Cells, Effector Memory Conv T Cells, Naive Conv T Cells and Stem Cell Memory-like Conv T Cells in iLN
Description: as for outcome 12
Time Frame: Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of total Conv T cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of total Conv T cells
  CD45RA+ Effector Memory Conv T cells | 1.14 (0.152) | 0.88 (0.180)
  Central Memory Conv T cells | 23.07 (2.646) | 25.03 (2.923)
  Effector Memory Conv T cells | 20.43 (2.422) | 18.28 (2.692)
  Naive Conv T cells | 46.13 (3.081) | 46.93 (3.454)
  Stem Cell Memory-like Conv T cells | 1.35 (0.176) | 1.57 (0.201)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.26, 95% CI [-0.23 to 0.75], Standard Error of Mean 0.236 — The mean difference in CD45RA+ Effector Memory Conv T cells (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -1.95, 95% CI 2-sided [-10.20 to 6.29], Standard Error of Mean 3.943 — The mean difference in Central Memory Conv T cells (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 2.15, 95% CI 2-sided [-5.38 to 9.69], Standard Error of Mean 3.621 — The mean difference in Effector Memory Conv T cells(Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 4: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.80, 95% CI 2-sided [-10.47 to 8.86], Standard Error of Mean 4.629 — The mean difference in Naive Conv T cells (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 5: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.77 to 0.34], Standard Error of Mean 0.268 — The mean difference in Stem cell Memory-like Conv T cells (Healthy participants versus NOT1D participants) in iLN has been presented

19. Primary Outcome: Percentage of Leukocyte Subsets Including TFH Cells, PD-1+ ICOS+ TFH Cells, Type 17 T Helper (TH17) Cells, TH1 Cells, TH1 TH17 Cells, TH1 TH17 TH2 T Cells, TH1 TH2 Cells, TH2 Cells, and TH22 Cells in Blood
Description: Peripheral blood samples were collected from both healthy and NOT1D participants at the indicated time points for the analysis of leukocyte subsets from T cell Panel. Candidate biomarkers associated with either location of cells and/or disease-status were identified using flow cytometry technique. Generalized linear mixed models were used to analyze data separately for each flow cytometry cell type to provide estimates for comparisons. Fixed categorical were group, sample type, and the interaction of group with sample type, where Group was HV or NOT1D, and sample type was peripheral blood, core biopsy or FNA. Only those participants with data available at specific time point were analyzed (represented by n=x in category titles).
Time Frame: Pre Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of total memory Conv T cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of total memory Conv T cells
  TFH cells; n=12, 10 | 16.77 (1.723) | 21.86 (1.888)
  PD-1+ ICOS+ TFH cells; n=6, 7: number analyzed (Participants) | 6 | 7
  PD-1+ ICOS+ TFH cells; n=6, 7 | 0.13 (0.036) | 0.18 (0.035)
  TH17 cells; n=12, 10 | 7.79 (0.963) | 7.89 (1.055)
  TH1 cells; n=12, 10 | 19.69 (2.895) | 17.60 (3.172)
  TH1 TH17 cells; n=12, 10 | 16.25 (1.606) | 16.22 (1.759)
  TH1 TH17 TH2 T cells; n=12, 10 | 7.16 (0.750) | 7.16 (0.821)
  TH1 TH2 cells; n=12, 10 | 9.30 (0.692) | 9.90 (0.758)
  TH2 cells; n=12, 10 | 8.46 (0.994) | 6.89 (1.089)
  TH22 cells; n=12, 10 | 3.00 (0.340) | 3.01 (0.372)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -5.09, 95% CI 2-sided [-10.42 to 0.25], Standard Error of Mean 2.556 — The mean difference in TFH cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.15 to 0.07], Standard Error of Mean 0.050 — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-3.08 to 2.88], Standard Error of Mean 1.428 — The mean difference in TH17 cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 4: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 2.09, 95% CI 2-sided [-6.87 to 11.05], Standard Error of Mean 4.294 — The mean difference in TH1 cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 5: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-4.94 to 5.00], Standard Error of Mean 2.382 — The mean difference in TH1 TH17 cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 6: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-2.31 to 2.32], Standard Error of Mean 1.112 — The mean difference in TH1 TH17 TH2 T cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 7: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.59, 95% CI 2-sided [-2.73 to 1.55], Standard Error of Mean 1.026 — The mean difference in TH1 TH2 cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 8: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 1.57, 95% CI 2-sided [-1.51 to 4.64], Standard Error of Mean 1.474 — The mean difference in TH2 cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 9: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-1.05 to 1.05], Standard Error of Mean 0.504 — The mean difference in TH22 cells (Healthy participants versus NOT1D participants) in blood has been presented

20. Primary Outcome: Percentage of Leukocyte Subsets Including TFH Cells, PD-1+ ICOS+ TFH Cells, Type 17 T Helper (TH17) Cells, TH1 Cells, TH1 TH17 Cells, TH1 TH17 TH2 T Cells, TH1 TH2 Cells, TH2 Cells, and TH22 Cells in iLN
Description: Samples were collected including up to two FNA passages of iLN and up to five core biopsies of iLN at the indicated time point from both healthy and NOT1D participants for the analysis of leukocyte subsets from T cell Panel. Candidate biomarkers associated with either location of cells and/or disease-status were identified using flow cytometry technique. Generalized linear mixed models were used to analyze data separately for each flow cytometry cell type to provide estimates for comparisons. Fixed categorical were group, sample type, and the interaction of group with sample type, where Group was HV or NOT1D, and sample type was peripheral blood, core biopsy or FNA. Only those participants with data available at specific time point were analyzed (represented by n=x in category titles).
Time Frame: Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percenatge of total memory Conv T cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percenatge of total memory Conv T cells
  TFH cells; n=12,10 | 23.02 (2.385) | 21.48 (2.706)
  PD-1+ ICOS+ TFH cells; n=10,10: number analyzed (Participants) | 10 | 10
  PD-1+ ICOS+ TFH cells; n=10,10 | 1.30 (0.662) | 1.93 (0.542)
  TH17 cells; n=12,10 | 6.56 (0.932) | 6.15 (1.033)
  TH1 cells; n=12,10 | 15.08 (1.878) | 18.58 (2.110)
  TH1 TH17 cells; n=11,10: number analyzed (Participants) | 11 | 10
  TH1 TH17 cells; n=11,10 | 3.03 (0.483) | 2.78 (0.558)
  TH1 TH17 TH2 T cells; n=11,10: number analyzed (Participants) | 11 | 10
  TH1 TH17 TH2 T cells; n=11,10 | 1.94 (0.360) | 1.54 (0.409)
  TH1 TH2 cells; n=12,10 | 7.73 (0.816) | 7.25 (0.942)
  TH2 cells; n=12,10 | 20.03 (1.754) | 16.98 (1.975)
  TH22 cells; n=12,10 | 1.50 (0.277) | 1.48 (0.352)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 1.54, 95% CI 2-sided [-5.99 to 9.07], Standard Error of Mean 3.607 — The mean difference in TFH cells (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-2.43 to 1.18], Standard Error of Mean 0.855 — The mean difference in PD-1+ ICOS+ TFH cells (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.41, 95% CI 2-sided [-2.49 to 3.31], Standard Error of Mean 1.391 — The mean difference in TH17 cells (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 4: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -3.50, 95% CI 2-sided [-9.39 to 2.39], Standard Error of Mean 2.824 — The mean difference in TH1 cells (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 5: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-1.29 to 1.78], Standard Error of Mean 0.738 — The mean difference in TH1 TH17 cells (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 6: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.40, 95% CI 2-sided [-0.73 to 1.54], Standard Error of Mean 0.544 — The mean difference in TH1 TH17 TH2 T cells (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 7: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.48, 95% CI 2-sided [-2.12 to 3.07], Standard Error of Mean 1.246 — The mean difference in TH1 TH2 cells (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 8: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 3.05, 95% CI 2-sided [-2.45 to 8.55], Standard Error of Mean 2.641 — The mean difference in TH2 cells (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 9: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.92 to 0.96], Standard Error of Mean 0.448 — The mean difference in TH22 cells (Healthy participants versus NOT1D participants) in iLN has been presented

21. Primary Outcome: Percentage of Leukocyte Subsets Including TFH Cells, PD-1+ ICOS+ TFH Cells, TH1 Cells, TH1 TH17 Cells, TH1 TH17 TH2 Cells, TH1 TH2 Cells, TH17 Cells, TH2 Cells and TH22 Cells-like Reg T Cells in Blood
Description: Peripheral blood samples were collected from both healthy and NOT1D participants at the indicated time points for the analysis of leukocyte subsets from T cell Panel. Candidate biomarkers associated with either location of cells and/or disease-status were identified using flow cytometry technique. Generalized linear mixed models were used to analyze data separately for each flow cytometry cell type to provide estimates for comparisons. Fixed categorical were group, sample type, and the interaction of group with sample type, where Group was HV or NOT1D, and sample type was peripheral blood, core biopsy or FNA. NA indicates that data was not availble. Only those participants with data available at specific time point were analyzed (represented by n=x in category titles).
Time Frame: Pre Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of total memory Reg T cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of total memory Reg T cells
  TFH cells-like Reg T cells; n=12, 10 | 11.63 (1.901) | 16.46 (2.083)
  PD-1+ ICOS+ TFH cells-like Reg T cells; n=0, 0: number analyzed (Participants) | 0 | 0
  TH1 cells-like Reg T cells; n=12, 10 | 5.35 (0.643) | 6.18 (0.704)
  TH1 TH17-like Reg T cells; n=7, 7: number analyzed (Participants) | 7 | 7
  TH1 TH17-like Reg T cells; n=7, 7 | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis. | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.
  TH1 TH17 TH2 cells-like Reg T cells; n=12, 10 | 10.48 (1.036) | 13.36 (1.135)
  TH1 TH2 cells-like Reg T cells; n=12, 10 | 12.04 (0.649) | 10.24 (0.711)
  TH17 cells-like Reg T cells; n=12, 10 | 17.37 (0.869) | 17.67 (0.952)
  TH2 cells-like Reg T cells; n=12, 10 | 12.47 (1.285) | 9.09 (1.408)
  TH22 cells-like Reg T cells; n=12, 10 | 11.46 (0.953) | 12.63 (1.044)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -4.83, 95% CI 2-sided [-10.71 to 1.05], Standard Error of Mean 2.820 — The mean difference in TFH cells-like Reg T cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-2.82 to 1.16], Standard Error of Mean 0.953 — The mean difference in TH1 cells-like Reg T cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -2.88, 95% CI [-6.08 to 0.33], Standard Error of Mean 1.536 — The mean difference in TH1 TH17 TH2 cells-like Reg T cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 4: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 1.81, 95% CI 2-sided [-0.20 to 3.81], Standard Error of Mean 0.963 — The mean difference in TH1 TH2 cells-like Reg T cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 5: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-2.99 to 2.39], Standard Error of Mean 1.289 — The mean difference in TH17 cells-like Reg T cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 6: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 3.38, 95% CI 2-sided [-0.59 to 7.36], Standard Error of Mean 1.907 — The mean difference in TH2 cells-like Reg T cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 7: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -1.16, 95% CI 2-sided [-4.11 to 1.78], Standard Error of Mean 1.413 — The mean difference in TH22 cells-like Reg T cells (Healthy participants versus NOT1D participants) in blood has been presented

22. Primary Outcome: Percentage of Leukocyte Subsets Including TFH Cells, PD-1+ ICOS+ TFH Cells, TH1 Cells, TH1 TH17 Cells, TH1 TH17 TH2 Cells, TH1 TH2 Cells, TH17 Cells, TH2 Cells and TH22 Cells-like Reg T Cells in iLN
Description: Samples were collected including up to two FNA passages of iLN and up to five core biopsies of iLN at the indicated time point from both healthy and NOT1D participants for the analysis of leukocyte subsets from T cell Panel. Candidate biomarkers associated with either location of cells and/or disease-status were identified using flow cytometry technique. Generalized linear mixed models were used to analyze data separately for each flow cytometry cell type to provide estimates for comparisons. Fixed categorical were group, sample type, and the interaction of group with sample type, where Group was HV or NOT1D, and sample type was peripheral blood, core biopsy or FNA. Only those participants with data available at specific time point were analyzed (represented by n=x in category titles). NA indicates that data was not available.
Time Frame: Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of total memory Reg T cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of total memory Reg T cells
  TFH cells-like Reg T cells; n=12, 10 | 13.48 (1.913) | 12.97 (2.203)
  PD-1+ ICOS+ TFH cells-like Reg T cells; n=5,7: number analyzed (Participants) | 5 | 7
  PD-1+ ICOS+ TFH cells-like Reg T cells; n=5,7 | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis. | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.
  TH1 cells-like Reg T cells; n=12, 10 | 7.31 (1.202) | 11.41 (1.395)
  TH1 TH17-like Reg T cells; n=1, 2: number analyzed (Participants) | 1 | 2
  TH1 TH17-like Reg T cells; n=1, 2 | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis. | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.
  TH1 TH17 TH2 cells-like Reg T cells; n=7, 6: number analyzed (Participants) | 7 | 6
  TH1 TH17 TH2 cells-like Reg T cells; n=7, 6 | 2.56 (0.839) | 4.11 (0.871)
  TH1 TH2 cells-like Reg T cells; n=12, 10 | 10.12 (1.085) | 10.99 (1.342)
  TH17 cells-like Reg T cells; n=12, 10 | 7.20 (1.418) | 7.67 (1.673)
  TH2 cells-like Reg T cells; n=12, 10 | 27.83 (2.262) | 27.24 (2.546)
  TH22 cells-like Reg T cells; n=8, 7: number analyzed (Participants) | 8 | 7
  TH22 cells-like Reg T cells; n=8, 7 | 2.29 (0.513) | 2.70 (0.628)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.51, 95% CI 2-sided [-5.60 to 6.63], Standard Error of Mean 2.918 — The mean difference in TFH cells-like Reg T cells (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -4.10, 95% CI 2-sided [-7.93 to -0.26], Standard Error of Mean 1.842 — The mean difference in TH1 cells-like Reg T cells (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -1.55, 95% CI 2-sided [-4.34 to 1.24], Standard Error of Mean 1.209 — The mean difference in TH1 TH17 TH2 cells-like Reg T cells (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 4: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.87, 95% CI 2-sided [-4.51 to 2.77], Standard Error of Mean 1.725 — The mean difference in TH1 TH2 cells-like Reg T cells (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 5: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-5.02 to 4.09], Standard Error of Mean 2.193 — The mean difference in TH17 cells-like Reg T cells (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 6: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.58, 95% CI 2-sided [-6.52 to 7.68], Standard Error of Mean 3.405 — The mean difference in TH2 cells-like Reg T cells (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 7: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-2.21 to 1.40], Standard Error of Mean 0.811 — The mean difference in TH22 cells-like Reg T cells (Healthy participants versus NOT1D participants) in iLN has been presented

23. Primary Outcome: Percentage of Leukocyte Subsets Including Reg T Cells in Blood
Description: Peripheral blood samples were collected from both healthy and NOT1D participants at the indicated time points for the analysis of leukocyte subsets from T Reg cell Panel. Candidate biomarkers associated with either location of cells and/or disease-status were identified using flow cytometry technique. Generalized linear mixed models were used to analyze data separately for each flow cytometry cell type to provide estimates for comparisons. Fixed categorical were group, sample type, and the interaction of group with sample type, where Group was HV or NOT1D, and sample type was peripheral blood, core biopsy or FNA.
Time Frame: Pre Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of CD4 T cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of CD4 T cells | 6.95 (0.405) | 6.56 (0.444)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.40, 95% CI 2-sided [-0.86 to 1.65], Standard Error of Mean 0.601 — The mean difference in Reg T cells (Healthy participants versus NOT1D participants) in blood has been presented

24. Primary Outcome: Percentage of Leukocyte Subsets Including Reg T Cells in iLN
Description: Samples were collected including up to two FNA passages of iLN and up to five core biopsies of iLN at the indicated time point from both healthy and NOT1D participants for the analysis of leukocyte subsets from T Reg cell Panel. Candidate biomarkers associated with either location of cells and/or disease-status were identified using flow cytometry technique. Generalized linear mixed models were used to analyze data separately for each flow cytometry cell type to provide estimates for comparisons. Fixed categorical were group, sample type, and the interaction of group with sample type, where Group was HV or NOT1D, and sample type was peripheral blood, core biopsy or FNA.
Time Frame: Biopsy session on Day 1
Population: Safety Population. Only those participants with data available at specified time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of CD4 T cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 11 | 9
Percentage of CD4 T cells | 12.04 (0.631) | 12.28 (0.682)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-2.18 to 1.70], Standard Error of Mean 0.929 — The mean difference in Reg T cells (Healthy participants versus NOT1D participants) in iLN has been presented

25. Primary Outcome: Percentage of Leukocyte Subsets Including CD69+ CD8 and Antigen Ki67 (Ki67)+ CD8 in Blood
Description: as for outcome 23
Time Frame: Pre Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of CD8 T cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of CD8 T cells
  CD69+ CD8 cells | 3.23 (0.299) | 2.28 (0.327)
  Ki67+ CD8 cells | 1.06 (0.391) | 1.89 (0.429)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.95, 95% CI 2-sided [0.02 to 1.87], Standard Error of Mean 0.443 — The mean difference in CD69+ CD8 cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-2.04 to 0.38], Standard Error of Mean 0.580 — The mean difference in Ki67+ CD8 cells (Healthy participants versus NOT1D participants) in blood has been presented

26. Primary Outcome: Percentage of Leukocyte Subsets Including CD69+ CD8 and Antigen Ki67 (Ki67)+ CD8 in iLN
Description: Samples were collected including up to two FNA passages of iLN and up to five core biopsies of iLN at the indicated time point from both healthy and NOT1D participants for the analysis of leukocyte subsets from T Reg cell Panel. Candidate biomarkers associated with either location of cells and/or disease-status were identified using flow cytometry technique. Generalized linear mixed models were used to analyze data separately for each flow cytometry cell type to provide estimates for comparisons. Fixed categorical were group, sample type, and the interaction of group with sample type, where Group was HV or NOT1D, and sample type was peripheral blood, core biopsy or FNA. Only those participants with data available at specific time point were analyzed (represented by n=x in category titles).
Time Frame: Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of CD8 T cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of CD8 T cells
  CD69+ CD8 cells; n=11, 9: number analyzed (Participants) | 11 | 9
  CD69+ CD8 cells; n=11, 9 | 17.77 (2.950) | 20.54 (3.127)
  Ki67+ CD8 cells; n= 11, 6: number analyzed (Participants) | 11 | 6
  Ki67+ CD8 cells; n= 11, 6 | 5.86 (0.646) | 3.66 (0.828)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -2.77, 95% CI 2-sided [-11.81 to 6.27], Standard Error of Mean 4.299 — The mean difference in CD69+ CD8 cells (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 2.20, 95% CI 2-sided [-0.04 to 4.44], Standard Error of Mean 1.051 — The mean difference in Ki67+ CD8 cells (Healthy participants versus NOT1D participants) in iLN has been presented

27. Primary Outcome: Percentage of Leukocyte Subsets Including CD15s+ Reg T Cells, CD69+ Reg T Cells, Helios+ Reg T Cells, Ki67+ T Reg Cells, Memory Reg T Cells and Resting Reg T Cells in Blood
Description: Peripheral blood samples were collected from both healthy and NOT1D participants at the indicated time points for the analysis of leukocyte subsets from T Reg cell Panel. Candidate biomarkers associated with either location of cells and/or disease-status were identified using flow cytometry technique. Generalized linear mixed models were used to analyze data separately for each flow cytometry cell type to provide estimates for comparisons. Fixed categorical were group, sample type, and the interaction of group with sample type, where Group was HV or NOT1D, and sample type was peripheral blood, core biopsy or FNA. Only those participants with data available at specific time point were analyzed (represented by n=x in category titles).
Time Frame: Pre Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of T Reg cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of T Reg cells
  CD15s+ Reg T cells; n= 12, 10 | 7.84 (1.492) | 9.13 (1.635)
  CD69+ Reg T cells; n= 11, 10: number analyzed (Participants) | 11 | 10
  CD69+ Reg T cells; n= 11, 10 | 3.19 (0.213) | 2.27 (0.223)
  Helios+ Reg T cells; n= 12, 10 | 75.19 (2.034) | 70.98 (2.228)
  Ki67+ T Reg cells; n= 12, 10 | 5.34 (0.664) | 6.32 (0.727)
  Memory Reg T cells; n= 12, 10 | 40.93 (2.563) | 45.79 (2.808)
  Resting Reg T cells n= 12, 10 | 45.34 (3.191) | 36.74 (3.496)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -1.29, 95% CI 2-sided [-5.91 to 3.32], Standard Error of Mean 2.214 — The mean difference in CD15s+ Reg T cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.92, 95% CI 2-sided [0.28 to 1.57], Standard Error of Mean 0.308 — The mean difference in CD69+ Reg T cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 4.21, 95% CI 2-sided [-2.08 to 10.51], Standard Error of Mean 3.017 — The mean difference in Helios+ Reg T cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 4: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.98, 95% CI 2-sided [-3.03 to 1.08], Standard Error of Mean 0.985 — The mean difference in Ki67+ T Reg cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 5: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -4.86, 95% CI 2-sided [-12.80 to 3.07], Standard Error of Mean 3.802 — The mean difference in Memory Reg T cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 6: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 8.60, 95% CI 2-sided [-1.27 to 18.47], Standard Error of Mean 4.733 — The mean difference in Resting Reg T cells (Healthy participants versus NOT1D participants) in blood has been presented

28. Primary Outcome: Percentage of Leukocyte Subsets Including CD15s+ Reg T Cells, CD69+ Reg T Cells, Helios+ Reg T Cells, Ki67+ T Reg Cells, Memory Reg T Cells and Resting Reg T Cells in iLN
Description: as for outcome 26
Time Frame: Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of T Reg cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of T Reg cells
  CD15s+ Reg T cells; n=11, 8: number analyzed (Participants) | 11 | 8
  CD15s+ Reg T cells; n=11, 8 | 16.54 (3.248) | 10.01 (3.675)
  CD69+ Reg T cells; n= 11, 9: number analyzed (Participants) | 11 | 9
  CD69+ Reg T cells; n= 11, 9 | 48.02 (3.034) | 56.55 (3.451)
  Helios+ Reg T cells; n=11,9: number analyzed (Participants) | 11 | 9
  Helios+ Reg T cells; n=11,9 | 81.28 (1.723) | 79.17 (1.837)
  Ki67+ T Reg cell; n= 10, 8: number analyzed (Participants) | 10 | 8
  Ki67+ T Reg cell; n= 10, 8 | 8.39 (1.347) | 5.09 (1.505)
  Memory Reg T cells; n= 11, 9: number analyzed (Participants) | 11 | 9
  Memory Reg T cells; n= 11, 9 | 50.12 (2.660) | 49.90 (3.022)
  Resting Reg T cells; n=11,9: number analyzed (Participants) | 11 | 9
  Resting Reg T cells; n=11,9 | 35.32 (3.031) | 27.00 (3.453)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 6.53, 95% CI [-3.78 to 16.85], Standard Error of Mean 4.905 — The mean difference in CD15s+ Reg T cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -8.54, 95% CI 2-sided [-18.17 to 1.10], Standard Error of Mean 4.595 — The mean difference in CD69+ Reg T cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 2.11, 95% CI 2-sided [-3.23 to 7.45], Standard Error of Mean 2.519 — The mean difference in Helios+ Reg T cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 4: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 3.30, 95% CI 2-sided [-0.98 to 7.59], Standard Error of Mean 2.020 — The mean difference in Ki67+ T Reg cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 5: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-8.23 to 8.67], Standard Error of Mean 4.026 — The mean difference in Memory Reg T cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 6: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 8.31, 95% CI 2-sided [-1.32 to 17.95], Standard Error of Mean 4.595 — The mean difference in Resting Reg T cells (Healthy participants versus NOT1D participants) in blood has been presented

29. Primary Outcome: Percentage of Leukocyte Subsets Including CD15s+ Conv T Cells, CD69+ Conv T Cells, Helios+ Conv T Cells and Ki67+ Conv T Cells in Blood
Description: as for outcome 23
Time Frame: Pre Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of total Conv T cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of total Conv T cells
  CD15s+ Conv T cells | 2.59 (0.405) | 2.28 (0.444)
  CD69+ Conv T cells | 2.05 (0.206) | 1.41 (0.226)
  Helios+ Conv T cells | 2.07 (0.233) | 1.68 (0.255)
  Ki67+ Conv T cells | 1.02 (0.202) | 1.18 (0.221)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.32, 95% CI 2-sided [-0.94 to 1.57], Standard Error of Mean 0.601 — The mean difference in CD15s+ Conv T cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.64, 95% CI 2-sided [0.00 to 1.28], Standard Error of Mean 0.306 — The mean difference in CD69+ Conv T cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.39, 95% CI 2-sided [-0.33 to 1.11], Standard Error of Mean 0.345 — The mean difference in Helios+ Conv T cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 4: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.78 to 0.47], Standard Error of Mean 0.300 — The mean difference in Ki67+ Conv T cells (Healthy participants versus NOT1D participants) in blood has been presented

30. Primary Outcome: Percentage of Leukocyte Subsets Including CD15s+ Conv T Cells, CD69+ Conv T Cells, Helios+ Conv T Cells and Ki67+ Conv T Cells in iLN
Description: as for outcome 26
Time Frame: Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of total Conv T cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of total Conv T cells
  CD15s+ Conv T cells; n=11, 8: number analyzed (Participants) | 11 | 8
  CD15s+ Conv T cells; n=11, 8 | 4.43 (0.653) | 2.65 (0.743)
  CD69+ Conv T cells; n=11, 9: number analyzed (Participants) | 11 | 9
  CD69+ Conv T cells; n=11, 9 | 27.74 (3.060) | 30.29 (3.589)
  Helios+ Conv T cells;n=11,9: number analyzed (Participants) | 11 | 9
  Helios+ Conv T cells;n=11,9 | 5.50 (0.631) | 5.35 (0.720)
  Ki67+ Conv T cells; n= 11,8: number analyzed (Participants) | 11 | 8
  Ki67+ Conv T cells; n= 11,8 | 4.39 (0.560) | 1.65 (0.669)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 1.78, 95% CI 2-sided [-0.30 to 3.86], Standard Error of Mean 0.989 — The mean difference in CD15s+ Conv T cells (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -2.55, 95% CI 2-sided [-12.45 to 7.35], Standard Error of Mean 4.716 — The mean difference in CD69+ Conv T cells (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-1.86 to 2.14], Standard Error of Mean 0.957 — The mean difference in Helios+ Conv T cells (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 4: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 2.74, 95% CI 2-sided [0.90 to 4.58], Standard Error of Mean 0.872 — The mean difference in Ki67+ Conv T cells (Healthy participants versus NOT1D participants) in iLN has been presented

31. Primary Outcome: Percentage of Leukocyte Subsets Including CD15s+ Memory Conv T Cells, CD69+ Memory Conv T Cells, Helios+ Memory Conv T Cells and Ki67+ Memory Conv T Cells in Blood
Description: as for outcome 23
Time Frame: Pre Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of total memory Conv T cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of total memory Conv T cells
  CD15s+ Memory Conv T cells | 5.39 (0.906) | 4.82 (0.993)
  CD69+ Memory Conv T cells | 2.53 (0.237) | 1.69 (0.259)
  Helios+ Memory Conv T cells | 3.46 (0.401) | 2.64 (0.439)
  Ki67+ Memory Conv T cells | 2.03 (0.397) | 2.34 (0.435)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.57, 95% CI 2-sided [-2.23 to 3.38], Standard Error of Mean 1.344 — The mean difference in CD15s+ Memory Conv T cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.84, 95% CI 2-sided [0.10 to 1.57], Standard Error of Mean 0.351 — The mean difference in CD69+ Memory Conv T cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.83, 95% CI 2-sided [-0.41 to 2.07], Standard Error of Mean 0.594 — The mean difference in Helios+ Memory Conv T cells (Healthy participants versus NOT1D participants) in blood has been presented
Statistical Analysis 4: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-1.54 to 0.92], Standard Error of Mean 0.589 — The mean difference in Ki67+ Memory Conv T cells (Healthy participants versus NOT1D participants) in blood has been presented

32. Primary Outcome: Percentage of Leukocyte Subsets Including CD15s+ Memory Conv T Cells, CD69+ Memory Conv T Cells, Helios+ Memory Conv T Cells and Ki67+ Memory Conv T Cells in iLN
Description: as for outcome 26
Time Frame: Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of total memory Conv T cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of total memory Conv T cells
  CD15s+ Memory Conv T cells; n=11, 8: number analyzed (Participants) | 11 | 8
  CD15s+ Memory Conv T cells; n=11, 8 | 7.60 (1.131) | 4.59 (1.307)
  CD69+ Memory Conv T cells; n=11, 9: number analyzed (Participants) | 11 | 9
  CD69+ Memory Conv T cells; n=11, 9 | 44.32 (2.739) | 46.38 (3.433)
  Helios+ Memory Conv T cells; n= 11, 9: number analyzed (Participants) | 11 | 9
  Helios+ Memory Conv T cells; n= 11, 9 | 8.25 (1.450) | 6.97 (1.438)
  Ki67+ Memory Conv T cells; n=11,8: number analyzed (Participants) | 11 | 8
  Ki67+ Memory Conv T cells; n=11,8 | 4.47 (0.545) | 2.33 (0.643)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 3.01, 95% CI 2-sided [-0.62 to 6.63], Standard Error of Mean 1.728 — The mean difference in CD15s+ Memory Conv T cells (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -2.06, 95% CI 2-sided [-11.33 to 7.21], Standard Error of Mean 4.392 — The mean difference in CD69+ Memory Conv T cells (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 1.28, 95% CI 2-sided [-14.56 to 17.13], Standard Error of Mean 2.042 — The mean difference in Helios+ Memory Conv T cells (Healthy participants versus NOT1D participants) in iLN has been presented
Statistical Analysis 4: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 2.14, 95% CI 2-sided [0.36 to 3.92], Standard Error of Mean 0.843 — The mean difference in Ki67+ Memory Conv T cells (Healthy participants versus NOT1D participants) in iLN has been presented

33. Secondary Outcome: Percentage of Leukocyte Subsets Including B Lymphocytes, Classical B Lymphocytes, Double Negative B Lymphocytes, Naive B Lymphocytes, Plasmablast and Transitional B Lymphocytes in iLN Core Biopsies and iLN FNA
Description: as for outcome 2
Time Frame: Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of B lymphocytes
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of B lymphocytes
  Circulating B Lymphocytes; FNA; n=9,4: number analyzed (Participants) | 9 | 4
  Circulating B Lymphocytes; FNA; n=9,4 | 14.36 (2.104) | 12.07 (2.272)
  Circulating B Lymphocytes; Core; n=4, 8: number analyzed (Participants) | 4 | 8
  Circulating B Lymphocytes; Core; n=4, 8 | 16.66 (1.668) | 12.20 (1.633)
  Classical B Lymphocytes; FNA; n=9,4: number analyzed (Participants) | 9 | 4
  Classical B Lymphocytes; FNA; n=9,4 | 39.89 (4.438) | 28.35 (6.283)
  Classical B Lymphocytes; Core; n= 4, 8: number analyzed (Participants) | 4 | 8
  Classical B Lymphocytes; Core; n= 4, 8 | 37.66 (4.711) | 32.02 (3.716)
  Double Negative B Lymphocytes; FNA; n=9,4: number analyzed (Participants) | 9 | 4
  Double Negative B Lymphocytes; FNA; n=9,4 | 8.48 (2.285) | 9.85 (2.430)
  Double Negative B Lymphocytes; Core; n= 4, 8: number analyzed (Participants) | 4 | 8
  Double Negative B Lymphocytes; Core; n= 4, 8 | 8.89 (1.302) | 10.68 (1.177)
  Naive B Lymphocytes;FNA; n=9,4: number analyzed (Participants) | 9 | 4
  Naive B Lymphocytes;FNA; n=9,4 | 36.05 (3.545) | 44.36 (4.939)
  Naive B Lymphocytes; Core; n= 4, 8: number analyzed (Participants) | 4 | 8
  Naive B Lymphocytes; Core; n= 4, 8 | 35.60 (4.671) | 43.91 (3.796)
  Plasmablast; FNA; n=4, 3: number analyzed (Participants) | 4 | 3
  Plasmablast; FNA; n=4, 3 | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis. | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.
  Plasmablast; Core; n=0, 5: number analyzed (Participants) | 0 | 5
  Plasmablast; Core; n=0, 5 |  | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.
  Transitional B Lymphocytes; FNA; n=2, 1: number analyzed (Participants) | 2 | 1
  Transitional B Lymphocytes; FNA; n=2, 1 | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis. | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.
  Transitional B Lymphocytes;Core; n=1, 2: number analyzed (Participants) | 1 | 2
  Transitional B Lymphocytes;Core; n=1, 2 | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis. | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 2.29, 95% CI 2-sided [-4.24 to 8.83], Standard Error of Mean 3.097 — The mean difference in Circulating B Lymphocytes (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 4.46, 95% CI 2-sided [-0.47 to 9.39], Standard Error of Mean 2.334 — The mean difference in Circulating B Lymphocytes (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 11.54, 95% CI 2-sided [-5.24 to 28.32], Standard Error of Mean 7.693 — The mean difference in Classical B Lymphocytes (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 4: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 5.64, 95% CI 2-sided [-7.73 to 19.01], Standard Error of Mean 6.000 — The mean difference in Classical B Lymphocytes (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 5: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -1.37, 95% CI 2-sided [-8.46 to 5.71], Standard Error of Mean 3.336 — The mean difference in Double Negative B Lymphocytes (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 6: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -1.78, 95% CI 2-sided [-5.54 to 1.98], Standard Error of Mean 1.755 — The mean difference in Double Negative B Lymphocytes (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 7: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -8.30, 95% CI 2-sided [-21.58 to 4.98], Standard Error of Mean 6.080 — The mean difference in Naive B Lymphocytes (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 8: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -8.31, 95% CI 2-sided [-21.49 to 4.87], Standard Error of Mean 6.019 — The mean difference in Naive B Lymphocytes by (Healthy participants versus NOT1D participants) core biopsy method has been presented

34. Secondary Outcome: Percentage of Leukocyte Subsets Including B-cells, CD56+ CD16+, CD56bright NK Cells, CD56lo CD16+, CD56lo CD16, Dendritic Cells, NK Cells in iLN Core Biopsies and iLN FNA
Description: as for outcome 2
Time Frame: Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of mononuclear cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of mononuclear cells
  B-cells; FNA; n=9, 4: number analyzed (Participants) | 9 | 4
  B-cells; FNA; n=9, 4 | 10.48 (1.417) | 5.51 (2.106)
  B-cells; Core; n=4, 8: number analyzed (Participants) | 4 | 8
  B-cells; Core; n=4, 8 | 7.29 (2.411) | 9.17 (1.769)
  CD56+CD16+; FNA; n=8, 2: number analyzed (Participants) | 8 | 2
  CD56+CD16+; FNA; n=8, 2 | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis. | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.
  CD56+CD16+; Core; n=2, 7: number analyzed (Participants) | 2 | 7
  CD56+CD16+; Core; n=2, 7 | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis. | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.
  CD56bright NK cells; FNA; n=9, 4: number analyzed (Participants) | 9 | 4
  CD56bright NK cells; FNA; n=9, 4 | 0.61 (0.110) | 0.47 (0.154)
  CD56bright NK cells; Core; n=4, 8: number analyzed (Participants) | 4 | 8
  CD56bright NK cells; Core; n=4, 8 | 0.47 (0.118) | 0.53 (0.089)
  CD56lo CD16+; FNA; n=9, 4: number analyzed (Participants) | 9 | 4
  CD56lo CD16+; FNA; n=9, 4 | 0.55 (0.215) | 0.94 (0.340)
  CD56lo CD16+; Core; n=3, 8: number analyzed (Participants) | 3 | 8
  CD56lo CD16+; Core; n=3, 8 | 0.82 (0.272) | 0.45 (0.152)
  CD56lo CD16-; FNA; n=8, 4: number analyzed (Participants) | 8 | 4
  CD56lo CD16-; FNA; n=8, 4 | 0.19 (0.042) | 0.21 (0.053)
  CD56lo CD16-; Core; n=3,7: number analyzed (Participants) | 3 | 7
  CD56lo CD16-; Core; n=3,7 | 0.18 (0.054) | 0.21 (0.041)
  Dendritic cells; FNA; n=9, 4: number analyzed (Participants) | 9 | 4
  Dendritic cells; FNA; n=9, 4 | 0.47 (0.061) | 0.24 (0.097)
  Dendritic cells; Core; n=4, 8: number analyzed (Participants) | 4 | 8
  Dendritic cells; Core; n=4, 8 | 0.44 (0.183) | 0.54 (0.125)
  NK cells; FNA; n=9, 4: number analyzed (Participants) | 9 | 4
  NK cells; FNA; n=9, 4 | 1.60 (0.425) | 1.66 (0.637)
  NK cells; Core; n=4, 8: number analyzed (Participants) | 4 | 8
  NK cells; Core; n=4, 8 | 1.27 (0.333) | 1.35 (0.251)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 4.97, 95% CI 2-sided [-0.54 to 10.48], Standard Error of Mean 2.538 — The mean difference in B-cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -1.88, 95% CI 2-sided [-8.37 to 4.61], Standard Error of Mean 2.990 — The mean difference in B-cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.26 to 0.54], Standard Error of Mean 0.189 — The mean difference in CD56bright NK cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 4: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.37 to 0.27], Standard Error of Mean 0.147 — The mean difference in CD56bright NK cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 5: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-1.27 to 0.49], Standard Error of Mean 0.402 — The mean difference in CD56lo CD16+ (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 6: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.37, 95% CI 2-sided [-0.33 to 1.07], Standard Error of Mean 0.312 — The mean difference in CD56lo CD16+ (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 7: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.16 to 0.13], Standard Error of Mean 0.068 — The mean difference in CD56lo CD16- by (Healthy participants versus NOT1D participants) FNA method has been presented
Statistical Analysis 8: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.17 to 0.12], Standard Error of Mean 0.068 — The mean difference in CD56lo CD16- (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 9: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-0.03 to 0.47], Standard Error of Mean 0.114 — The mean difference in Dendritic cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 10: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.59 to 0.40], Standard Error of Mean 0.221 — The mean difference in Dendritic cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 11: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-1.72 to 1.60], Standard Error of Mean 0.766 — The mean difference in NK cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 12: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.99 to 0.82], Standard Error of Mean 0.417 — The mean difference in NK cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented

35. Secondary Outcome: Percentage of Leukocyte Subsets Including CD56+CD16+, CD56br NK Cells CD56lo CD16+ and CD56lo CD16- in iLN Core Biopsies and iLN FNA
Description: as for outcome 2
Time Frame: Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of NK cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of NK cells
  CD56+CD16+; FNA; n=8, 2: number analyzed (Participants) | 8 | 2
  CD56+CD16+; FNA; n=8, 2 | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis. | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.
  CD56+CD16+; Core; n=2, 7: number analyzed (Participants) | 2 | 7
  CD56+CD16+; Core; n=2, 7 | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis. | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.
  CD56bright NK cells; FNA; n=9, 4: number analyzed (Participants) | 9 | 4
  CD56bright NK cells; FNA; n=9, 4 | 40.37 (3.934) | 26.65 (6.356)
  CD56bright NK cells; Core; n=4, 8: number analyzed (Participants) | 4 | 8
  CD56bright NK cells; Core; n=4, 8 | 43.32 (6.340) | 43.36 (4.129)
  CD56lo CD16+; FNA; n=9, 4: number analyzed (Participants) | 9 | 4
  CD56lo CD16+; FNA; n=9, 4 | 34.66 (4.476) | 54.69 (7.327)
  CD56lo CD16+; Core; n=3, 8: number analyzed (Participants) | 3 | 8
  CD56lo CD16+; Core; n=3, 8 | 39.58 (11.072) | 35.32 (6.300)
  CD56lo CD16-; FNA; n=8, 4: number analyzed (Participants) | 8 | 4
  CD56lo CD16-; FNA; n=8, 4 | 13.17 (1.321) | 13.31 (2.039)
  CD56lo CD16-; Core; n=3, 7: number analyzed (Participants) | 3 | 7
  CD56lo CD16-; Core; n=3, 7 | 12.42 (3.479) | 15.21 (2.258)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 13.72, 95% CI 2-sided [-2.72 to 30.15], Standard Error of Mean 7.475 — [estimate comment as in outcome 34, analysis 3]
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-16.85 to 16.78], Standard Error of Mean 7.566 — [estimate comment as in outcome 34, analysis 4]
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -20.03, 95% CI 2-sided [-38.98 to -1.08], Standard Error of Mean 8.586 — The mean difference in CD56lo CD16+ (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 4: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 4.25, 95% CI 2-sided [-24.14 to 32.65], Standard Error of Mean 12.739 — The mean difference in CD56lo CD16+ by (Healthy participants versus NOT1D participants) core biopsy method has been presented
Statistical Analysis 5: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-5.54 to 5.26], Standard Error of Mean 2.429 — The mean difference in CD56lo CD16- (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 6: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -2.79, 95% CI 2-sided [-12.31 to 6.73], Standard Error of Mean 4.148 — [estimate comment as in outcome 34, analysis 8]

36. Secondary Outcome: Percentage of Leukocyte Subsets Including Myeloid Dendritic Cells and Plasmacytoid Dendritic Cells in iLN Core Biopsies and iLN FNA
Description: Samples were collected including up to two FNA passages of iLN and up to five core biopsies of iLN at the indicated time point from both healthy and NOT1D participants for the analysis of leukocyte subsets from Monocyte Panel. Candidate biomarkers associated with either location of cells and/or disease-status were identified using flow cytometry technique. Generalized linear mixed models were used to analyze data separately for each flow cytometry cell type to provide estimates for comparisons. Fixed categorical were group, sample type, and the interaction of group with sample type, where Group was HV or NOT1D, and sample type was peripheral blood, core biopsy or FNA. Only those participants with data available at specific time point were analyzed (represented by n=x in category titles).
Time Frame: Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of total dendritic cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of total dendritic cells
  Myeloid Dendritic cells; FNA; n=8, 4: number analyzed (Participants) | 8 | 4
  Myeloid Dendritic cells; FNA; n=8, 4 | 46.76 (4.383) | 38.50 (6.298)
  Myeloid Dendritic cells; Core; n=4 ,8: number analyzed (Participants) | 4 | 8
  Myeloid Dendritic cells; Core; n=4 ,8 | 39.16 (4.626) | 22.95 (4.111)
  Plasmacytoid Dendritic cells; FNA; n=9, 3: number analyzed (Participants) | 9 | 3
  Plasmacytoid Dendritic cells; FNA; n=9, 3 | 54.59 (5.834) | 62.48 (8.742)
  Plasmacytoid Dendritic cells; Core; n=4, 8: number analyzed (Participants) | 4 | 8
  Plasmacytoid Dendritic cells; Core; n=4, 8 | 60.27 (4.185) | 74.12 (3.988)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 8.25, 95% CI 2-sided [-8.58 to 25.08], Standard Error of Mean 7.673 — The mean difference in Myeloid Dendritic cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 16.22, 95% CI 2-sided [3.17 to 29.26], Standard Error of Mean 6.189 — The mean difference in Myeloid Dendritic cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -7.89, 95% CI 2-sided [-31.03 to 15.25], Standard Error of Mean 10.509 — The mean difference in Plasmacytoid Dendritic cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 4: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -13.85, 95% CI 2-sided [-26.04 to -1.66], Standard Error of Mean 5.781 — The mean difference in (Healthy participants versus NOT1D participants) by core biopsy method has been presented

37. Secondary Outcome: Percentage of Leukocyte Subsets Including CD14+ CD16+ Monocytes, CD14+ Monocytes and CD16+ Monocytes in iLN Core Biopsies and iLN FNA
Description: Samples were collected including up to two FNA passages of iLN and up to five core biopsies of iLN at the indicated time point from both healthy and NOT1D participants for the analysis of leukocyte subsets from Monocyte Panel. Candidate biomarkers associated with either location of cells and/or disease-status were identified using flow cytometry technique. Only those participants with data available at specific time point were analyzed (represented by n=x in category titles). NA indicates data was not available.
Time Frame: Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of monocytes
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of monocytes
  CD14+ CD16+ monocytes; ;FNA; n=0, 1: number analyzed (Participants) | 0 | 1
  CD14+ CD16+ monocytes; ;FNA; n=0, 1 |  | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.
  CD14+ CD16+ monocytes; Core; n=0, 0: number analyzed (Participants) | 0 | 0
  CD14+ monocytes; ;FNA; n=5, 2: number analyzed (Participants) | 5 | 2
  CD14+ monocytes; ;FNA; n=5, 2 | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis. | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.
  CD14+ monocytes;Core; n=3, 3: number analyzed (Participants) | 3 | 3
  CD14+ monocytes;Core; n=3, 3 | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis. | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.
  CD16+ monocytes; ;FNA; n=0, 2: number analyzed (Participants) | 0 | 2
  CD16+ monocytes; ;FNA; n=0, 2 |  | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.
  CD16+ monocytes; ;FNA; n=0,0: number analyzed (Participants) | 0 | 0

38. Secondary Outcome: Percentage of Leukocyte Subsets Including CD45RA+ Effector Memory CD8, Central Memory CD8, Effector Memory CD8, Naive CD8 and Stem Cell Memory-like CD8 in iLN Core Biopsies and iLN FNA
Description: as for outcome 20
Time Frame: Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of CD8 T cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of CD8 T cells
  CD45RA+ Effector Memory CD8; FNA; n=12, 8: number analyzed (Participants) | 12 | 8
  CD45RA+ Effector Memory CD8; FNA; n=12, 8 | 11.96 (2.298) | 13.58 (2.721)
  CD45RA+ Effector Memory CD8; Core; n=11, 10: number analyzed (Participants) | 11 | 10
  CD45RA+ Effector Memory CD8; Core; n=11, 10 | 17.12 (2.342) | 13.11 (2.489)
  Central Memory CD8; FNA; n=12, 7: number analyzed (Participants) | 12 | 7
  Central Memory CD8; FNA; n=12, 7 | 4.84 (0.895) | 5.00 (1.113)
  Central Memory CD8; Core; n=11, 10: number analyzed (Participants) | 11 | 10
  Central Memory CD8; Core; n=11, 10 | 6.25 (1.264) | 7.41 (1.352)
  Effector Memory CD8; FNA; n=12, 8: number analyzed (Participants) | 12 | 8
  Effector Memory CD8; FNA; n=12, 8 | 11.32 (2.026) | 13.43 (2.389)
  Effector Memory CD8; Core; n= 11, 10: number analyzed (Participants) | 11 | 10
  Effector Memory CD8; Core; n= 11, 10 | 16.16 (2.105) | 17.76 (2.236)
  Naive CD8; FNA; n=12, 8: number analyzed (Participants) | 12 | 8
  Naive CD8; FNA; n=12, 8 | 61.17 (4.306) | 57.65 (4.994)
  Naive CD8; Core; n=11, 10: number analyzed (Participants) | 11 | 10
  Naive CD8; Core; n=11, 10 | 49.07 (4.888) | 51.25 (5.224)
  Stem Cell Memory-like CD8;FNA; n= 12, 6: number analyzed (Participants) | 12 | 6
  Stem Cell Memory-like CD8;FNA; n= 12, 6 | 1.73 (0.428) | 2.65 (0.563)
  Stem Cell Memory-like CD8; Core; 9,10: number analyzed (Participants) | 9 | 10
  Stem Cell Memory-like CD8; Core; 9,10 | 1.64 (0.257) | 2.06 (0.269)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -1.62, 95% CI 2-sided [-9.05 to 5.82], Standard Error of Mean 3.561 — The mean difference in CD45RA+ Effector Memory CD8 cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 4.01, 95% CI 2-sided [-3.13 to 11.16], Standard Error of Mean 3.418 — The mean difference in CD45RA+ Effector Memory CD8 cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-3.14 to 2.82], Standard Error of Mean 1.428 — The mean difference in Central Memory CD8 cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 4: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -1.16, 95% CI 2-sided [-5.03 to 2.71], Standard Error of Mean 1.851 — The mean difference in Central Memory CD8 cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 5: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -2.11, 95% CI 2-sided [-8.65 to 4.43], Standard Error of Mean 3.132 — The mean difference in Effector Memory CD8 cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 6: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -1.59, 95% CI 2-sided [-8.00 to 4.81], Standard Error of Mean 3.071 — The mean difference in Effector Memory CD8 cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 7: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 3.51, 95% CI 2-sided [-10.21 to 17.24], Standard Error of Mean 6.594 — The mean difference in Naive CD8 cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 8: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -2.18, 95% CI 2-sided [-17.10 to 12.74], Standard Error of Mean 7.155 — The mean difference in Naive CD8 cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 9: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.92, 95% CI 2-sided [-2.42 to 0.58], Standard Error of Mean 0.708 — The mean difference in Stem Cell Memory-like CD8 cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 10: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-1.19 to 0.35], Standard Error of Mean 0.372 — The mean difference in Stem Cell Memory-like CD8 cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented

39. Secondary Outcome: Percentage of Leukocyte Subsets Including PD-1+ ICOS+ TFH Cell-like Reg T Cells in iLN Core Biopsies and iLN FNA
Description: Samples were collected including up to two FNA passages of iLN and up to five core biopsies of iLN at the indicated time point from both healthy and NOT1D participants for the analysis of leukocyte subsets from T cell Panel. Candidate biomarkers associated with either location of cells and/or disease-status were identified using flow cytometry technique. Only those participants with data available at specific time point were analyzed (represented by n=x in category titles). NA indicates that data was not available.
Time Frame: Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of TFH cell-like Reg T Cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of TFH cell-like Reg T Cells
  PD-1+ ICOS+ TFH cell-like Reg T cells; FNA;n=2, 3: number analyzed (Participants) | 2 | 3
  PD-1+ ICOS+ TFH cell-like Reg T cells; FNA;n=2, 3 | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis. | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.
  PD-1+ ICOS+ TFH cell-like Reg T cells; Core; n=4,5: number analyzed (Participants) | 4 | 5
  PD-1+ ICOS+ TFH cell-like Reg T cells; Core; n=4,5 | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis. | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.

40. Secondary Outcome: Percentage of Leukocyte Subsets Including PD-1+ ICOS+ TFH Cells in iLN Core Biopsies and iLN FNA
Description: as for outcome 20
Time Frame: Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of TFH cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of TFH cells
  PD-1+ ICOS+ TFH cells; FNA; n=8, 4: number analyzed (Participants) | 8 | 4
  PD-1+ ICOS+ TFH cells; FNA; n=8, 4 | 3.95 (1.601) | 9.34 (1.977)
  PD-1+ ICOS+ TFH cells; Core; n=6, 10: number analyzed (Participants) | 6 | 10
  PD-1+ ICOS+ TFH cells; Core; n=6, 10 | 1.55 (5.416) | 8.58 (4.613)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -5.39, 95% CI 2-sided [-11.56 to 0.78], Standard Error of Mean 2.545 — The mean difference in PD-1+ ICOS+ TFH cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -7.03, 95% CI 2-sided [-22.22 to 8.16], Standard Error of Mean 7.114 — The mean difference in PD-1+ ICOS+ TFH cells (Healthy participants versus NOT1D participants) by core biopsy FNA method has been presented

41. Secondary Outcome: Percentage of Leukocyte Subsets Including Central Memory Conv T Cells, Effector Memory Conv T Cells, Naive Conv T Cells and Stem Cell Memory-like Conv T Cells in iLN Core Biopsies and iLN FNA
Description: as for outcome 20
Time Frame: Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of total Conv T cell
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of total Conv T cell
  CD45RA+ Effector Memory Conv T cells; FNA; n=12, 7: number analyzed (Participants) | 12 | 7
  CD45RA+ Effector Memory Conv T cells; FNA; n=12, 7 | 1.16 (0.221) | 0.77 (0.282)
  CD45RA+ Effector Memory Conv T cells;Core;n=11, 10: number analyzed (Participants) | 11 | 10
  CD45RA+ Effector Memory Conv T cells;Core;n=11, 10 | 1.13 (0.126) | 0.99 (0.133)
  Central Memory Conv T cells; FNA; n= 12, 8: number analyzed (Participants) | 12 | 8
  Central Memory Conv T cells; FNA; n= 12, 8 | 21.15 (2.765) | 21.34 (3.188)
  Central Memory Conv T cells; Core; n= 11, 10: number analyzed (Participants) | 11 | 10
  Central Memory Conv T cells; Core; n= 11, 10 | 24.99 (2.881) | 28.71 (3.087)
  Effector Memory Conv T cells; FNA; n=12, 8: number analyzed (Participants) | 12 | 8
  Effector Memory Conv T cells; FNA; n=12, 8 | 17.71 (2.605) | 15.46 (3.080)
  Effector Memory Conv T cells; Core; n=11, 10: number analyzed (Participants) | 11 | 10
  Effector Memory Conv T cells; Core; n=11, 10 | 23.16 (2.736) | 21.10 (2.909)
  Naive Conv T cells; FNA; n=12,8: number analyzed (Participants) | 12 | 8
  Naive Conv T cells; FNA; n=12,8 | 50.43 (3.672) | 52.52 (4.395)
  Naive Conv T cells; Core; n=11, 10: number analyzed (Participants) | 11 | 10
  Naive Conv T cells; Core; n=11, 10 | 41.82 (3.421) | 41.34 (3.614)
  Stem Cell Memory-like Conv T cells; FNA; n=12, 7: number analyzed (Participants) | 12 | 7
  Stem Cell Memory-like Conv T cells; FNA; n=12, 7 | 1.39 (0.191) | 1.40 (0.249)
  Stem Cell Memory-like Conv T cells; Core; n=11, 10: number analyzed (Participants) | 11 | 10
  Stem Cell Memory-like Conv T cells; Core; n=11, 10 | 1.31 (0.224) | 1.73 (0.236)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.39, 95% CI 2-sided [-0.36 to 1.14], Standard Error of Mean 0.358 — The mean difference in CD45RA+ Effector Memory Conv T cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.25 to 0.52], Standard Error of Mean 0.184 — The mean difference in CD45RA+ Effector Memory Conv T cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-9.02 to 8.64], Standard Error of Mean 4.220 — The mean difference in Central Memory Conv T cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 4: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -3.72, 95% CI 2-sided [-12.57 to 5.13], Standard Error of Mean 4.223 — The mean difference in Central Memory Conv T cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 5: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 2.25, 95% CI 2-sided [-6.16 to 10.66], Standard Error of Mean 4.034 — The mean difference in Effector Memory Conv T cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 6: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 2.06, 95% CI 2-sided [-6.27 to 10.39], Standard Error of Mean 3.994 — The mean difference in Effector Memory Conv T cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 7: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -2.09, 95% CI 2-sided [-14.09 to 9.92], Standard Error of Mean 5.727 — The mean difference in Naive Conv T cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 8: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.48, 95% CI 2-sided [-9.91 to 10.87], Standard Error of Mean 4.976 — The mean difference in Naive Conv T cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 9: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.67 to 0.65], Standard Error of Mean 0.314 — The mean difference in Stem Cell Memory-like Conv T cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 10: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-1.10 to 0.26], Standard Error of Mean 0.325 — The mean difference in Stem Cell Memory-like Conv T cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented

42. Secondary Outcome: Percentage of Leukocyte Subsets Including TFH Cells, PD-1+ ICOS+ TFH Cells, TH17 Cells, TH1 Cells, TH1 TH17 Cells, TH1 TH17 TH2 T Cells, TH1 TH2 Cells, TH2 Cells, and TH22 Cells in iLN Core Biopsies and iLN FNA
Description: as for outcome 20
Time Frame: Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percenatge of total memory Conv T cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percenatge of total memory Conv T cells
  TFH cells; ; FNA; n=12, 8: number analyzed (Participants) | 12 | 8
  TFH cells; ; FNA; n=12, 8 | 24.09 (2.913) | 17.09 (3.651)
  TFH cells; Core; n=11,10: number analyzed (Participants) | 11 | 10
  TFH cells; Core; n=11,10 | 21.94 (3.335) | 25.86 (3.491)
  PD-1+ ICOS+ TFH cells; FNA; n=8,4: number analyzed (Participants) | 8 | 4
  PD-1+ ICOS+ TFH cells; FNA; n=8,4 | 0.89 (0.356) | 2.15 (0.545)
  PD-1+ ICOS+ TFH cells; Core; n=6,10: number analyzed (Participants) | 6 | 10
  PD-1+ ICOS+ TFH cells; Core; n=6,10 | 1.72 (1.239) | 1.71 (0.859)
  TH17 cells;FNA; n=12,8: number analyzed (Participants) | 12 | 8
  TH17 cells;FNA; n=12,8 | 7.73 (1.122) | 6.96 (1.289)
  TH17 cells; Core; n=11,10: number analyzed (Participants) | 11 | 10
  TH17 cells; Core; n=11,10 | 5.38 (0.915) | 5.33 (0.977)
  TH1 cells; FNA; n=12,8: number analyzed (Participants) | 12 | 8
  TH1 cells; FNA; n=12,8 | 14.08 (2.340) | 15.05 (2.777)
  TH1 cells; Core; n=11,10: number analyzed (Participants) | 11 | 10
  TH1 cells; Core; n=11,10 | 16.09 (1.858) | 22.12 (1.970)
  TH1 TH17 cells; FNA; n=10,4: number analyzed (Participants) | 10 | 4
  TH1 TH17 cells; FNA; n=10,4 | 2.97 (0.510) | 3.07 (0.728)
  TH1 TH17 cells; Core; n=10,10: number analyzed (Participants) | 10 | 10
  TH1 TH17 cells; Core; n=10,10 | 3.08 (0.553) | 2.49 (0.559)
  TH1 TH17 TH2 T cells; FNA; n=10,4: number analyzed (Participants) | 10 | 4
  TH1 TH17 TH2 T cells; FNA; n=10,4 | 1.87 (0.371) | 1.44 (0.488)
  TH1 TH17 TH2 T cells; Core; n=10,10: number analyzed (Participants) | 10 | 10
  TH1 TH17 TH2 T cells; Core; n=10,10 | 2.01 (0.390) | 1.63 (0.409)
  TH1 TH2 cells; FNA; n=12,6: number analyzed (Participants) | 12 | 6
  TH1 TH2 cells; FNA; n=12,6 | 6.20 (0.910) | 5.68 (1.250)
  TH1 TH2 cells; Core; n=10, 10: number analyzed (Participants) | 10 | 10
  TH1 TH2 cells; Core; n=10, 10 | 9.25 (1.130) | 8.83 (1.147)
  TH2 cells; FNA; n=12,8: number analyzed (Participants) | 12 | 8
  TH2 cells; FNA; n=12,8 | 20.82 (2.168) | 18.67 (2.562)
  TH2 cells; Core; n=11,10: number analyzed (Participants) | 11 | 10
  TH2 cells; Core; n=11,10 | 19.24 (1.685) | 15.29 (1.821)
  TH22 cells; FNA; n=12,4: number analyzed (Participants) | 12 | 4
  TH22 cells; FNA; n=12,4 | 1.51 (0.336) | 1.46 (0.530)
  TH22 cells; Core; n=10, 10: number analyzed (Participants) | 10 | 10
  TH22 cells; Core; n=10, 10 | 1.49 (0.308) | 1.50 (0.311)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 7.00, 95% CI 2-sided [-2.80 to 16.81], Standard Error of Mean 4.671 — The mean difference in TFH cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -3.93, 95% CI 2-sided [-14.02 to 6.17], Standard Error of Mean 4.828 — The mean difference in TFH cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -1.26, 95% CI 2-sided [-2.69 to 0.16], Standard Error of Mean 0.651 — [estimate comment as in outcome 40, analysis 1]
Statistical Analysis 4: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-3.21 to 3.24], Standard Error of Mean 1.507 — The mean difference in PD-1+ ICOS+ TFH cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 5: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.77, 95% CI 2-sided [-2.78 to 4.33], Standard Error of Mean 1.709 — The mean difference in TH17 cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 6: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-2.75 to 2.85], Standard Error of Mean 1.339 — The mean difference in TH17 cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 7: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.97, 95% CI 2-sided [-8.56 to 6.63], Standard Error of Mean 3.631 — The mean difference in TH1 cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 8: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -6.03, 95% CI 2-sided [-11.69 to -0.38], Standard Error of Mean 2.708 — The mean difference in TH1 cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 9: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-1.98 to 1.78], Standard Error of Mean 0.889 — The mean difference in TH1 TH17 cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 10: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.59, 95% CI 2-sided [-1.07 to 2.24], Standard Error of Mean 0.787 — The mean difference in TH1 TH17 cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 11: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.43, 95% CI 2-sided [-0.85 to 1.72], Standard Error of Mean 0.613 — The mean difference in TH1 TH17 TH2 T cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 12: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [-0.80 to 1.56], Standard Error of Mean 0.565 — The mean difference in TH1 TH17 TH2 T cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 13: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.53, 95% CI 2-sided [-2.71 to 3.76], Standard Error of Mean 1.546 — The mean difference in TH1 TH2 cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 14: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.42, 95% CI 2-sided [-2.95 to 3.79], Standard Error of Mean 1.610 — The mean difference in TH1 TH2 cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 15: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 2.15, 95% CI 2-sided [-4.84 to 9.14], Standard Error of Mean 3.356 — The mean difference in TH2 cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 16: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 3.95, 95% CI 2-sided [-1.25 to 9.15], Standard Error of Mean 2.481 — The mean difference in TH2 cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 17: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-1.28 to 1.38], Standard Error of Mean 0.627 — The mean difference in TH22 cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 18: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.93 to 0.91], Standard Error of Mean 0.438 — The mean difference in TH22 cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented

43. Secondary Outcome: Percentage of Leukocyte Subsets Including TFH Cells, PD-1+ ICOS+ TFH Cells, TH1 Cells, TH1 TH17 Cells, TH1 TH17 TH2 Cells, TH1 TH2 Cells, TH17 Cells, TH2 Cells and TH22 Cells-like Reg T Cells in iLN Core Biopsies and iLN FNA
Description: as for outcome 22
Time Frame: Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of total memory Reg T cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of total memory Reg T cells
  TFH cells-like Reg T cells; FNA; n=11, 5: number analyzed (Participants) | 11 | 5
  TFH cells-like Reg T cells; FNA; n=11, 5 | 13.52 (2.224) | 13.22 (2.869)
  TFH cells-like Reg T cells; Core; n=9, 10: number analyzed (Participants) | 9 | 10
  TFH cells-like Reg T cells; Core; n=9, 10 | 13.44 (1.884) | 12.71 (1.926)
  PD-1+ ICOS+ TFH cells-like Reg T cells;FNA;n=2,3: number analyzed (Participants) | 2 | 3
  PD-1+ ICOS+ TFH cells-like Reg T cells;FNA;n=2,3 | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis. | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.
  PD-1+ ICOS+ TFH cells-like Reg T cells;Core;n=4,5: number analyzed (Participants) | 4 | 5
  PD-1+ ICOS+ TFH cells-like Reg T cells;Core;n=4,5 | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis. | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.
  TH1 cells-like Reg T cells;FNA; n=11,5: number analyzed (Participants) | 11 | 5
  TH1 cells-like Reg T cells;FNA; n=11,5 | 7.19 (1.428) | 12.09 (1.900)
  TH1 cells-like Reg T cells;Core;n=8, 10: number analyzed (Participants) | 8 | 10
  TH1 cells-like Reg T cells;Core;n=8, 10 | 7.43 (1.211) | 10.72 (1.167)
  TH1 TH17-like Reg T cells;FNA; n=1, 1: number analyzed (Participants) | 1 | 1
  TH1 TH17-like Reg T cells;FNA; n=1, 1 | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis. | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.
  TH1 TH17-like Reg T cells;Core; n=0,2: number analyzed (Participants) | 0 | 2
  TH1 TH17-like Reg T cells;Core; n=0,2 |  | NA (NA) — NA indicates that data was not available as the cell yield was too low to allow the analysis.
  TH1 TH17 TH2 cells-like Reg T cells;FNA; n=7, 4: number analyzed (Participants) | 7 | 4
  TH1 TH17 TH2 cells-like Reg T cells;FNA; n=7, 4 | 2.88 (0.599) | 3.17 (0.845)
  TH1 TH17 TH2 cells-like Reg T cells;Core;n=5,5: number analyzed (Participants) | 5 | 5
  TH1 TH17 TH2 cells-like Reg T cells;Core;n=5,5 | 2.25 (1.381) | 5.05 (1.348)
  TH1 TH2 cells-like Reg T cells;FNA; n=11, 4: number analyzed (Participants) | 11 | 4
  TH1 TH2 cells-like Reg T cells;FNA; n=11, 4 | 9.08 (1.092) | 10.52 (1.813)
  TH1 TH2 cells-like Reg T cells;Core; n=10,10: number analyzed (Participants) | 10 | 10
  TH1 TH2 cells-like Reg T cells;Core; n=10,10 | 11.15 (1.434) | 11.45 (1.460)
  TH17 cells-like Reg T cells;FNA; n=11, 4: number analyzed (Participants) | 11 | 4
  TH17 cells-like Reg T cells;FNA; n=11, 4 | 8.18 (1.547) | 9.64 (2.146)
  TH17 cells-like Reg T cells;Core; n=10, 10: number analyzed (Participants) | 10 | 10
  TH17 cells-like Reg T cells;Core; n=10, 10 | 6.23 (1.507) | 5.70 (1.582)
  TH2 cells-like Reg T cells;FNA; n=12, 8: number analyzed (Participants) | 12 | 8
  TH2 cells-like Reg T cells;FNA; n=12, 8 | 27.38 (2.749) | 29.63 (3.305)
  TH2 cells-like Reg T cells;Core; n=11, 10: number analyzed (Participants) | 11 | 10
  TH2 cells-like Reg T cells;Core; n=11, 10 | 28.28 (2.386) | 24.86 (2.522)
  TH22 cells-like Reg T cells;FNA; n=6,3: number analyzed (Participants) | 6 | 3
  TH22 cells-like Reg T cells;FNA; n=6,3 | 2.30 (0.653) | 2.95 (0.950)
  TH22 cells-like Reg T cells;Core; n=7,7: number analyzed (Participants) | 7 | 7
  TH22 cells-like Reg T cells;Core; n=7,7 | 2.28 (0.619) | 2.45 (0.610)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.30, 95% CI 2-sided [-7.40 to 8.00], Standard Error of Mean 3.630 — The mean difference in TFH cells-like Reg T cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.72, 95% CI 2-sided [-4.90 to 6.35], Standard Error of Mean 2.694 — The mean difference in TFH cells-like Reg T cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -4.90, 95% CI 2-sided [-9.89 to 0.08], Standard Error of Mean 2.377 — The mean difference in TH1 cells-like Reg T cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 4: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -3.29, 95% CI 2-sided [-6.82 to 0.24], Standard Error of Mean 1.682 — The mean difference in TH1 cells-like Reg T cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 5: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-2.67 to 2.10], Standard Error of Mean 1.036 — The mean difference in TH1 TH17 TH2 cells-like Reg T cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 6: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -2.80, 95% CI 2-sided [-7.20 to 1.59], Standard Error of Mean 1.929 — The mean difference in TH1 TH17 TH2 cells-like Reg T cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 7: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -1.44, 95% CI 2-sided [-5.98 to 3.11], Standard Error of Mean 2.117 — The mean difference in TH1 TH2 cells-like Reg T cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 8: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-4.59 to 3.99], Standard Error of Mean 2.047 — The mean difference in TH1 TH2 cells-like Reg T cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 9: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -1.47, 95% CI 2-sided [-6.99 to 4.06], Standard Error of Mean 2.645 — The mean difference in TH17 cells-like Reg T cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 10: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.53, 95% CI 2-sided [-4.05 to 5.11], Standard Error of Mean 2.185 — The mean difference in TH17 cells-like Reg T cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 11: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -2.25, 95% CI 2-sided [-11.23 to 6.73], Standard Error of Mean 4.299 — The mean difference in TH2 cells-like Reg T cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 12: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 3.42, 95% CI 2-sided [-3.84 to 10.67], Standard Error of Mean 3.472 — The mean difference in TH2 cells-like Reg T cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 13: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.65, 95% CI 2-sided [-3.30 to 2.00], Standard Error of Mean 1.153 — The mean difference in TH22 cells-like Reg T cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 14: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-2.06 to 1.72], Standard Error of Mean 0.869 — The mean difference in TH22 cells-like Reg T cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented

44. Secondary Outcome: Percentage of Leukocyte Subsets Including Reg T Cells in iLN Core Biopsies and iLN FNA
Description: as for outcome 26
Time Frame: Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of CD4 T cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of CD4 T cells
  Reg T cells; FNA; n=10, 4: number analyzed (Participants) | 10 | 4
  Reg T cells; FNA; n=10, 4 | 11.98 (0.750) | 11.52 (1.067)
  Reg T cells; Core; n=5, 9: number analyzed (Participants) | 5 | 9
  Reg T cells; Core; n=5, 9 | 12.11 (0.871) | 13.05 (0.597)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.46, 95% CI 2-sided [-2.27 to 3.19], Standard Error of Mean 1.304 — The mean difference in Reg T cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.94, 95% CI 2-sided [-3.24 to 1.36], Standard Error of Mean 1.056 — The mean difference in Reg T cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented

45. Secondary Outcome: Percentage of Leukocyte Subsets Including CD69+ CD8 and Antigen Ki67 (Ki67)+ CD8 in iLN Core Biopsies and iLN FNA
Description: as for outcome 26
Time Frame: Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of CD8 T cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of CD8 T cells
  CD69+ CD8 cells; FNA; n=10, 4: number analyzed (Participants) | 10 | 4
  CD69+ CD8 cells; FNA; n=10, 4 | 16.80 (2.837) | 17.97 (4.201)
  CD69+ CD8 cells; Core; n=5, 9: number analyzed (Participants) | 5 | 9
  CD69+ CD8 cells; Core; n=5, 9 | 18.74 (4.287) | 23.12 (3.117)
  Ki67+ CD8 cells; FNA; n=9, 3: number analyzed (Participants) | 9 | 3
  Ki67+ CD8 cells; FNA; n=9, 3 | 4.82 (0.689) | 3.33 (1.189)
  Ki67+ CD8 cells; Core; n=4, 6: number analyzed (Participants) | 4 | 6
  Ki67+ CD8 cells; Core; n=4, 6 | 6.90 (1.025) | 3.99 (0.785)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -1.16, 95% CI 2-sided [-11.91 to 9.58], Standard Error of Mean 5.069 — The mean difference in CD69+ CD8 cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -4.38, 95% CI 2-sided [-15.85 to 7.10], Standard Error of Mean 5.301 — The mean difference in CD69+ CD8 cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 1.48, 95% CI 2-sided [-1.62 to 4.59], Standard Error of Mean 1.374 — The mean difference in Ki67+ CD8 cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 4: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 2.91, 95% CI 2-sided [-0.05 to 5.88], Standard Error of Mean 1.291 — The mean difference in Ki67+ CD8 cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented

46. Secondary Outcome: Percentage of Leukocyte Subsets Including CD15s+ Reg T Cells, CD69+ Reg T Cells, Helios+ Reg T Cells, Ki67+ T Reg Cells, Memory Reg T Cells and Resting Reg T Cells in iLN Core Biopsies and iLN FNA
Description: as for outcome 26
Time Frame: Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of T Reg cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of T Reg cells
  CD15s+ Reg T cells; FNA; n=9, 4: number analyzed (Participants) | 9 | 4
  CD15s+ Reg T cells; FNA; n=9, 4 | 12.99 (2.022) | 8.13 (2.327)
  CD15s+ Reg T cells; Core; n=4, 8: number analyzed (Participants) | 4 | 8
  CD15s+ Reg T cells; Core; n=4, 8 | 20.10 (4.531) | 11.89 (5.044)
  CD69+ Reg T cells; FNA; n=10, 4: number analyzed (Participants) | 10 | 4
  CD69+ Reg T cells; FNA; n=10, 4 | 48.55 (3.666) | 59.74 (4.510)
  CD69+ Reg T cells; Core; n=5, 9: number analyzed (Participants) | 5 | 9
  CD69+ Reg T cells; Core; n=5, 9 | 47.48 (2.744) | 53.37 (2.708)
  Helios+ Reg T cells; FNA; n=10, 4: number analyzed (Participants) | 10 | 4
  Helios+ Reg T cells; FNA; n=10, 4 | 80.88 (1.559) | 79.23 (1.929)
  Helios+ Reg T cells; Core; n=5, 9: number analyzed (Participants) | 5 | 9
  Helios+ Reg T cells; Core; n=5, 9 | 81.68 (2.180) | 79.10 (1.968)
  Ki67+ T Reg cells; FNA; n=8, 4: number analyzed (Participants) | 8 | 4
  Ki67+ T Reg cells; FNA; n=8, 4 | 8.02 (1.855) | 4.80 (2.072)
  Ki67+ T Reg cells; Core; n=4, 7: number analyzed (Participants) | 4 | 7
  Ki67+ T Reg cells; Core; n=4, 7 | 8.76 (0.893) | 5.38 (0.996)
  Memory Reg T cells; FNA; n=10, 4: number analyzed (Participants) | 10 | 4
  Memory Reg T cells; FNA; n=10, 4 | 47.10 (2.842) | 48.55 (3.788)
  Memory Reg T cells; Core; n=5, 9: number analyzed (Participants) | 5 | 9
  Memory Reg T cells; Core; n=5, 9 | 53.13 (3.036) | 51.25 (2.818)
  Resting Reg T cells; FNA; n=9, 4: number analyzed (Participants) | 9 | 4
  Resting Reg T cells; FNA; n=9, 4 | 38.09 (3.392) | 27.64 (4.692)
  Resting Reg T cells; Core; n=5, 9: number analyzed (Participants) | 5 | 9
  Resting Reg T cells; Core; n=5, 9 | 32.54 (3.828) | 26.37 (3.080)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 4.86, 95% CI 2-sided [-1.60 to 11.31], Standard Error of Mean 3.083 — The mean difference in CD15s+ Reg T cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 8.21, 95% CI 2-sided [-6.15 to 22.57], Standard Error of Mean 6.780 — The mean difference in CD15s+ Reg T cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -11.19, 95% CI 2-sided [-23.48 to 1.11], Standard Error of Mean 5.812 — The mean difference in CD69+ Reg T cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 4: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -5.89, 95% CI 2-sided [-14.14 to 2.37], Standard Error of Mean 3.855 — The mean difference in CD69+ Reg T cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 5: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 1.65, 95% CI 2-sided [-3.54 to 6.84], Standard Error of Mean 2.480 — The mean difference in Helios+ Reg T cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 6: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 2.57, 95% CI 2-sided [-3.84 to 8.98], Standard Error of Mean 2.937 — The mean difference in Helios+ Reg T cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 7: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 3.22, 95% CI 2-sided [-2.67 to 9.12], Standard Error of Mean 2.781 — The mean difference in Ki67+ T Reg cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 8: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 3.38, 95% CI 2-sided [0.55 to 6.21], Standard Error of Mean 1.337 — The mean difference in Ki67+ T Reg cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 9: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -1.45, 95% CI 2-sided [-11.49 to 8.58], Standard Error of Mean 4.736 — The mean difference in Memory Reg T cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 10: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 1.88, 95% CI 2-sided [-6.81 to 10.58], Standard Error of Mean 4.142 — The mean difference in Memory Reg T cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 11: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 10.45, 95% CI 2-sided [-2.01 to 22.92], Standard Error of Mean 5.790 — The mean difference in Resting Reg T cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 12: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 6.17, 95% CI 2-sided [-4.24 to 16.59], Standard Error of Mean 4.913 — The mean difference in Resting Reg T cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented

47. Secondary Outcome: Percentage of Leukocyte Subsets Including CD15s+ Conv T Cells, CD69+ Conv T Cells, Helios+ Conv T Cells and Ki67+ Conv T Cells in iLN Core Biopsies and iLN FNA
Description: as for outcome 26
Time Frame: Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of total Conv T cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of total Conv T cells
  CD15s+ Conv T cells;FNA;n=9, 4: number analyzed (Participants) | 9 | 4
  CD15s+ Conv T cells;FNA;n=9, 4 | 3.02 (0.448) | 1.64 (0.533)
  CD15s+ Conv T cells; Core; n=5, 8: number analyzed (Participants) | 5 | 8
  CD15s+ Conv T cells; Core; n=5, 8 | 5.85 (0.892) | 3.66 (0.978)
  CD69+ Conv T cells;FNA;n=10, 4: number analyzed (Participants) | 10 | 4
  CD69+ Conv T cells;FNA;n=10, 4 | 27.95 (3.498) | 28.86 (5.346)
  CD69+ Conv T cells; Core; n=5, 9: number analyzed (Participants) | 5 | 9
  CD69+ Conv T cells; Core; n=5, 9 | 27.54 (3.870) | 31.73 (2.943)
  Helios+ Conv T cells ; FNA;n=10, 4: number analyzed (Participants) | 10 | 4
  Helios+ Conv T cells ; FNA;n=10, 4 | 5.14 (0.750) | 5.27 (0.980)
  Helios+ Conv T cells ; Core; n=5, 9: number analyzed (Participants) | 5 | 9
  Helios+ Conv T cells ; Core; n=5, 9 | 5.85 (0.644) | 5.44 (0.570)
  Ki67+ Conv T cells; FNA;n=9, 4: number analyzed (Participants) | 9 | 4
  Ki67+ Conv T cells; FNA;n=9, 4 | 4.07 (0.760) | 0.86 (0.935)
  Ki67+ Conv T cells ; Core; n=5, 8: number analyzed (Participants) | 5 | 8
  Ki67+ Conv T cells ; Core; n=5, 8 | 4.72 (0.502) | 2.45 (0.505)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 1.38, 95% CI 2-sided [-0.08 to 2.83], Standard Error of Mean 0.696 — The mean difference in CD15s+ Conv T cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 2.19, 95% CI 2-sided [-0.61 to 4.98], Standard Error of Mean 1.324 — The mean difference in CD15s+ Conv T cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.91, 95% CI 2-sided [-14.66 to 12.85], Standard Error of Mean 6.389 — The mean difference in CD69+ Conv T cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 4: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -4.19, 95% CI 2-sided [-14.71 to 6.33], Standard Error of Mean 4.862 — The mean difference in CD69+ Conv T cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 5: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-2.73 to 2.47], Standard Error of Mean 1.234 — The mean difference in Helios+ Conv T cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 6: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 0.41, 95% CI 2-sided [-1.45 to 2.28], Standard Error of Mean 0.859 — The mean difference in Helios+ Conv T cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 7: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 3.21, 95% CI 2-sided [0.64 to 5.78], Standard Error of Mean 1.205 — The mean difference in Ki67+ Conv T cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 8: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 2.27, 95% CI 2-sided [0.75 to 3.79], Standard Error of Mean 0.712 — The mean difference in Ki67+ Conv T cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented

48. Secondary Outcome: Percentage of Leukocyte Subsets Including CD15s+ Memory Conv T Cells, CD69+ Memory Conv T Cells, Helios+ Memory Conv T Cells and Ki67+ Memory Conv T Cells in iLN Core Biopsies and iLN FNA
Description: as for outcome 26
Time Frame: Biopsy session on Day 1
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of total memory Conv cells
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Percentage of total memory Conv cells
  CD15s+ Memory Conv T cells; FNA; n=9, 4: number analyzed (Participants) | 9 | 4
  CD15s+ Memory Conv T cells; FNA; n=9, 4 | 6.39 (0.889) | 3.12 (1.042)
  CD15s+ Memory Conv T cells; Core; n=5, 8: number analyzed (Participants) | 5 | 8
  CD15s+ Memory Conv T cells; Core; n=5, 8 | 8.80 (1.390) | 6.06 (1.585)
  CD69+ Memory Conv T cells; FNA; n=10, 4: number analyzed (Participants) | 10 | 4
  CD69+ Memory Conv T cells; FNA; n=10, 4 | 45.74 (3.604) | 45.74 (5.662)
  CD69+ Memory Conv T cells; Core; n=5, 9: number analyzed (Participants) | 5 | 9
  CD69+ Memory Conv T cells; Core; n=5, 9 | 42.91 (3.198) | 47.03 (2.314)
  Helios+ Memory Conv T cells; FNA; n=9, 4: number analyzed (Participants) | 9 | 4
  Helios+ Memory Conv T cells; FNA; n=9, 4 | 7.68 (1.312) | 6.35 (2.661)
  Helios+ Memory Conv T cells; Core; n=5, 9: number analyzed (Participants) | 5 | 9
  Helios+ Memory Conv T cells; Core; n=5, 9 | 8.82 (2.144) | 7.59 (0.794)
  Ki67+ Memory Conv T cells; FNA; n=9, 4: number analyzed (Participants) | 9 | 4
  Ki67+ Memory Conv T cells; FNA; n=9, 4 | 4.32 (0.659) | 1.62 (0.777)
  Ki67+ Memory Conv T cells; Core; n=4, 8: number analyzed (Participants) | 4 | 8
  Ki67+ Memory Conv T cells; Core; n=4, 8 | 4.63 (0.482) | 3.04 (0.558)
Statistical Analysis 1: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 3.27, 95% CI 2-sided [0.40 to 6.15], Standard Error of Mean 1.370 — The mean difference in CD15s+ Memory Conv T cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 2: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 2.74, 95% CI 2-sided [-1.68 to 7.17], Standard Error of Mean 2.109 — The mean difference in CD15s+ Memory Conv T cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 3: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-14.49 to 14.48], Standard Error of Mean 6.712 — The mean difference in CD69+ Memory Conv T cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 4: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = -4.12, 95% CI 2-sided [-12.67 to 4.43], Standard Error of Mean 3.947 — The mean difference in CD69+ Memory Conv T cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 5: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 1.33, 95% CI 2-sided [-5.48 to 8.13], Standard Error of Mean 2.967 — The mean difference in Helios+ Memory Conv T cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 6: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 1.24, 95% CI 2-sided [-4.36 to 6.84], Standard Error of Mean 2.287 — The mean difference in Helios+ Memory Conv T cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented
Statistical Analysis 7: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 2.69, 95% CI 2-sided [0.54 to 4.84], Standard Error of Mean 1.019 — The mean difference in Ki67+ Memory Conv T cells (Healthy participants versus NOT1D participants) by FNA method has been presented
Statistical Analysis 8: Comparison: Healthy Participants vs Participants With NOT1D; Test type: Other; Mean Difference (Final Values) = 1.58, 95% CI 2-sided [0.03 to 3.13], Standard Error of Mean 0.737 — The mean difference in Ki67+ Memory Conv T cells (Healthy participants versus NOT1D participants) by core biopsy method has been presented

49. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Non-SAEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/ incapacity, is a congenital anomaly/ birth defect or other situations.
Time Frame: Up to Day 14
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Participants
  Any SAE | 0 | 0
  Any non-SAE | 9 | 5

50. Secondary Outcome: Number of Participants Undergoing Procedure Under Local Anesthetics
Description: Participants were asked to complete Pre-Biopsy Lymph Node Questionnaire about their expectations/experiences of undergoing the procedure of FNA biopsy followed by core needle biopsy. The number of participants who underwent procedure under local anesthetics have been presented.
Time Frame: Up to Day 4
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Participants | 6 | 7

51. Secondary Outcome: Number of Participants Undergoing iLN Biopsy Under Local Anesthetics
Description: Participants were asked to complete Pre-Biopsy Lymph Node Questionnaire about their expectations/experiences of undergoing the procedure of FNA biopsy followed by core needle biopsy. The number of participants who underwent iLN biopsy under local anesthetics have been presented.
Time Frame: Up to Day 4
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Participants | 0 | 0

52. Secondary Outcome: Number of Participants With Different Reasons for Participating in the Study
Description: Participants were asked to complete Pre-Biopsy Lymph Node Questionnaire about their expectations/experiences of undergoing the procedure of FNA biopsy followed by core needle biopsy. The different reasons have been listed as follows; have friend with diabetes mellitus (DM)/ to progress knowledge, to improve medicines development, participating in the study because of the honorarium, any other reason not listed above was categorized as "other" and participants having all three reasons as listed above to participate in the study were included in "All reasons" category
Time Frame: Up to Day 4
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Participants
  Have friend with DM/ to progress knowledge | 2 | 4
  To improve medicines development | 10 | 4
  Honorarium | 0 | 0
  Other | 0 | 1
  All reasons | 0 | 1

53. Secondary Outcome: Number of Participants With Extreme Anxiety Towards the Lymph Node Biopsy
Description: Participants were asked to complete Pre-Biopsy Lymph Node Questionnaire about their expectations/experiences of undergoing the procedure of FNA biopsy followed by core needle biopsy. The number of participants with extreme anxiety towards the procedure have been presented.
Time Frame: Up to Day 4
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Participants | 0 | 0

54. Secondary Outcome: Number of Participants Looking Forward to Undergo the Procedure
Description: Participants were asked to complete Pre-Biopsy Lymph Node Questionnaire about their expectations/experiences of undergoing the procedure of FNA biopsy followed by core needle biopsy. The number of participants looking forward to undergo the procedure have been presented.
Time Frame: Up to Day 4
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Participants | 1 | 0

55. Secondary Outcome: Number of Participants With Aspects Better Explained About the Lymph Node Biopsy Procedure
Description: Participants were asked to complete Post-Biopsy Lymph Node Questionnaire about their expectations/experiences of undergoing the procedure of FNA biopsy followed by core needle biopsy. The aspects better explained were as follows; itself, anesthetic procedure, after-care, none and any other procedure not listed above was categorized as "other".
Time Frame: Up to Day 4
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Participants
  Procedure itself | 1 | 1
  Anesthetic procedure | 0 | 0
  After-care | 1 | 0
  None | 9 | 9
  Other | 1 | 0

56. Secondary Outcome: Number of Participants Who Considered to Undergo Lymph Node Biopsy Procedure Another Time
Description: Participants were asked to complete Post-Biopsy Lymph Node Questionnaire about their expectations/experiences of undergoing the procedure of FNA biopsy followed by core needle biopsy. The number of participants who considered to undergo procedure another time have been presented.
Time Frame: Up to Day 4
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Participants | 10 | 9

57. Secondary Outcome: Number of Participants Who Were Encouraged to be Included in Study for iLN Biopsy
Description: Participants were asked to complete Post-Biopsy Lymph Node Questionnaire about their expectations/experiences of undergoing the procedure of FNA biopsy followed by core needle biopsy. Participants who were encouraged in study for iLN biopsy have been presented.
Time Frame: Up to Day 4
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Participants | 11 | 8

58. Secondary Outcome: Number of Participants Who Appreciated Receiving Study Feedback
Description: Participants were asked to complete Post-Biopsy Lymph Node Questionnaire about their expectations/experiences of undergoing the procedure of FNA biopsy followed by core needle biopsy. Participants who appreciated receiving study feedback have been presented.
Time Frame: Up to Day 4
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants | Participants With NOT1D
Number analyzed (Participants) | 12 | 10
Participants | 12 | 10

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (non-SAEs) were collected up to Day 14.
Description: SAEs and Non-SAEs were reported for Safety Population which comprised of all participants who completed any study assessment.
Arm/Group | Healthy Participants | Participants With NOT1D
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 9/12 | 5/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Participants (N=12) | Participants With NOT1D (N=10)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Post procedural contusion (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Procedural pain (Injury, poisoning and procedural complications) | 6 (6) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-03-06): https://cdn.clinicaltrials.gov/large-docs/42/NCT02801942/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-09): https://cdn.clinicaltrials.gov/large-docs/42/NCT02801942/SAP_001.pdf